CLINICAL TRIAL: NCT02725411
Title: A PHASE 3 RANDOMIZED, DOUBLE-BLIND, ACTIVE-CONTROLLED, MULTICENTER STUDY OF THE LONG-TERM SAFETY AND EFFICACY OF SUBCUTANEOUS ADMINISTRATION OF TANEZUMAB IN JAPANESE ADULT SUBJECTS WITH CHRONIC LOW BACK PAIN
Brief Title: Long Term Safety and Efficacy Study of Tanezumab in Japanese Adult Subjects With Chronic Low Back Pain
Acronym: TANGO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A4091063; JAPAN CLBP SC STUDY (Other: Alias Study Number)
Record Dates: First submitted 2016-01-20; First posted 2016-04-01 (Estimated); Results first posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-07

CONDITIONS: Low Back Pain
Keywords: Chronic low back pain; Chronic pain
MeSH Terms: conditions — Low Back Pain; Chronic Pain | interventions — Celecoxib; tanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Celecoxib (Active Comparator): Subcutaneous injection of placebo for tanezumab every 8 weeks plus oral celecoxib 100 mg twice daily for 56 weeks
  Interventions: Drug: Celecoxib; Biological: Placebo for tanezumab
- Tanezumab 5 mg (Experimental): Subcutaneous injection of tanezumab 5 mg every 8 weeks plus oral placebo for celecoxib twice daily for 56 weeks
  Interventions: Biological: Tanezumab 5 mg; Drug: Placebo for celecoxib
- Tanezumab 10 mg (Experimental): Subcutaneous injection of tanezumab 10 mg every 8 weeks plus oral placebo for celecoxib twice daily for 56 weeks
  Interventions: Biological: Tanezumab 10 mg; Drug: Placebo for celecoxib

INTERVENTIONS:
Drug: Celecoxib — Orally administered Celecoxib 100 mg twice daily for 56 weeks
  Arms: Celecoxib
Biological: Tanezumab 5 mg — Subcutaneous injection of tanezumab 5 mg every 8 weeks for 56 weeks
  Arms: Tanezumab 5 mg
Biological: Tanezumab 10 mg — Subcutaneous injection of tanezumab 10 mg every 8 weeks for 56 weeks
  Arms: Tanezumab 10 mg
Drug: Placebo for celecoxib — Orally administered the placebo twice daily for 56 weeks
  Arms: Tanezumab 10 mg; Tanezumab 5 mg
Biological: Placebo for tanezumab — Subcutaneous injection of the placebo every 8 weeks for 56 weeks
  Arms: Celecoxib

SUMMARY:
This study will investigate the long-term safety and efficacy of a fixed dose of tanezumab 5 mg and 10 mg administered subcutaneously (SC) seven times at 8 week intervals. The primary objective of this study is to evaluate the long term safety of tanezumab 5 mg and 10 mg administrated SC every 8 weeks (7 administrations). In addition, the study will evaluate the long term analgesic efficacy of tanezumab 5 mg and 10 mg SC administered every 8 weeks (7 administrations).

DETAILED DESCRIPTION:
This is a randomized, double-blind, active-controlled, multicenter, parallel-group Phase 3 study of the safety and efficacy of tanezumab when administered by SC injection for up to 56 weeks in subjects with chronic low back pain. Subjects will be randomized to 1 of 3 treatment groups in a 1:1:1 ratio. Treatment groups will include: 1) Placebo SC matching tanezumab administered at an 8-week interval (total of 7 times) plus celecoxib 100 mg twice a day (BID) to be administered orally for 56 weeks; 2) Tanezumab 5 mg SC administered at an 8-week interval (total of 7 times) plus placebo matching celecoxib to be administered orally BID for 56 weeks; 3) Tanezumab 10 mg SC administered at an 8-week interval (total of 7 times) plus placebo matching celecoxib to be administered orally BID for 56 weeks. The study is designed with a total duration (post-randomization) of up to 80 weeks and will consist of three periods: Screening (up to 37 days; includes a Washout Period and an Initial Pain Assessment Period [IPAP]), a Double-blind Treatment Period (56 weeks) and a Follow-up Period (24 weeks). The Screening Period (beginning up to 37 days prior to Randomization) includes a Washout Period (lasting 2 to 32 days), if required, and an IPAP (the 5 days prior to Randomization/Baseline). Prior to entering the study, subjects must be experiencing some benefit (eg, analgesic effect) from their current stable dose regimen of oral NSAID (celecoxib, loxoprofen or meloxicam) treatment, be tolerating their NSAID regimen, be taking this medication regularly (defined as an average of at least 5 days per week) during the 30 day period prior to the Screening Visit.

ELIGIBILITY:
Inclusion Criteria:

* Duration of chronic low back pain for ≥3 months, and treatment with agents for low back pain for ≥3 months.
* Primary location of low back pain must be between the 12th thoracic vertebra and the lower gluteal folds, with or without radiation into the posterior thigh, classified as Category 1 or 2 according to the classification of the Quebec Task Force in Spinal Disorders.
* Subjects must be experiencing some benefits from their current stable dose regimen of oral NSAID (celecoxib, loxoprofen or meloxicam) treatment as described in the protocol, be tolerating their NSAID regimen, be taking this medication regularly during the 30 day period prior to the Screening visit and must have had some improvement in low back pain, but still require additional pain relief at Screening.
* Subjects must maintain a stabilized, protocol specified NSAID dose regimen for at least the final 2 or 3 weeks of the Screening period.
* Low Back Pain Intensity (LBPI) score of ≥5 at Screening.
* Subjects must be willing to discontinue all pain medications for chronic low back pain except rescue medication and investigational product and not use prohibited pain medications throughout the duration of the study.
* Female subjects of childbearing potential and at risk for pregnancy must agree to comply with protocol specified contraceptive requirements.

Exclusion Criteria:

* Subjects exceeding protocol defined BMI limits.
* Diagnosis of osteoarthritis of the knee or hip as defined by the ACR combined clinical and radiographic criteria.

  * Subjects who have Kellgren Lawrence Grade > or =2 radiographic evidence of hip or Grade > or =3 radiographic evidence of knee osteoarthritis will be excluded.
  * Subjects who have Kellgren Lawrence Grade < or =2 radiographic evidence of knee osteoarthritis but who do not meet ACR criteria and do not have pain associated with their knee osteoarthritis will be allowed.
* Subjects with symptoms and radiologic findings consistent with osteoarthritis in the shoulder.
* History of lumbosacral radiculopathy within the past 2 years, history of spinal stenosis associated with neurological impairment, or history of neurogenic claudication.
* Back pain due to recent major trauma within 6 months prior to Screening.
* Surgical intervention during the past 6 months for the treatment of low back pain.
* Planned surgical procedure during the duration of the study.
* History or radiographic evidence of other diseases that could confound efficacy or safety assessments (eg, rheumatoid arthritis).
* History or radiographic evidence of orthopedic conditions that may increase the risk of, or confound assessment of joint safety conditions during the study.
* History of osteonecrosis or osteoporotic fracture.
* History of significant trauma or surgery to a knee, hip, or shoulder within the previous year.
* Signs or symptoms of carpal tunnel syndrome in the one year prior to Screening.
* Considered unfit for surgery based upon American Society of Anesthesiologists physical classification system for surgery grading, or subjects who would not be willing to undergo joint replacement surgery if required.
* History of intolerance or hypersensitivity to celecoxib/acetaminophen or any of its excipients or existence of a medical condition or use of concomitant medication for which the use of celecoxib/acetaminophen is contraindicated.
* Use of prohibited medications or prohibited non-pharmacological treatments without the appropriate washout period (if applicable) prior to Screening or IPAP.
* History of known alcohol, analgesic or narcotic abuse within 2 years of Screening.
* Presence of drugs of abuse or illegal drugs in the urine toxicology screen obtained at Screening.
* History of allergic or anaphylactic reaction to a therapeutic or diagnostic monoclonal antibody or IgG-fusion protein.
* Signs and symptoms of clinically significant cardiac disease.
* Poorly controlled hypertension as defined in the protocol or taking an antihypertensive that has not been stable for at least 1 month prior to Screening.
* Evidence of protocol defined orthostatic hypotension at Screening.
* Disqualifying score on the Survey of Autonomic Symptoms questionnaire at Screening.
* Diagnosis of a transient ischemic attack in the 6 months prior to Screening, diagnosis of stroke with residual deficits that would preclude completion of required study activities.
* History of cancer within 5 years prior to Screening, except for cutaneous basal cell or squamous cell cancer resolved by excision.
* Expected to undergo a therapeutic procedure or to use any analgesic other than those specified in the protocol throughout the pre-treatment and treatment periods that is likely to confound assessment of analgesic efficacy or safety.
* Previous exposure to exogenous NGF or to an anti-NGF antibody.
* Screening AST, ALT, serum creatinine or HbA1c values that exceed protocol defined limits.
* Positive Hepatitis B, Hepatitis C, or HIV tests at screening indicative of current infection.
* History, diagnosis, or signs and symptoms of clinically significant neurological disease or clinically significant psychiatric disorder.
* Pregnant, breastfeeding or female subjects of childbearing potential who are unwilling or unable to follow protocol required contraceptive requirements.
* Participation in other investigational drug studies within protocol defined time limits.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2016-05-26 (Actual); Primary Completion 2019-06-11 (Actual); Study Completion 2019-06-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (55):
- Japan (55):
  - Meitoh Hospital, Nagoya, Aichi-ken
  - Asahi Rosai Hospital, Owariasahi, Aichi-ken
  - Asahi General Hospital, Asahi, Chiba
  - Sato Orthopedic Clinic, Ichikawa, Chiba
  - Fukuoka Mirai Hospital, Higashi-ku,Fukuoka, Fukuoka
  - Shinkokura Hospital, Kitakyushu, Fukuoka
  - Kyushu Rosai Hospital, Kokuraminami-ku,Kitakyushu, Fukuoka
  - Kurume University Hospital, Kurume, Fukuoka
  - Shin Komonji Hospital, Moji-ku, Kitakyusyu, Fukuoka
  - Fujita general Hospital, Date-gun, Fukushima
  - Shirakawa Hospital, Shirakawa, Fukushima
  - Toyooka Chuo Hospital, Asahikawa, Hokkaido
  - Hakodate Central General Hospital, Hakodate, Hokkaido
  - Hakodate Ohmura Orthopedic Hospital, Hakodate, Hokkaido
  - Okubo Hospital, Akashi, Hyōgo
  - Omuro Orthopedic Clinic, Himeji, Hyōgo
  - Medical corporate corporation hoshikai Onishi medical clinic, Kako-gun, Hyōgo
  - Kobe Red Cross Hospital, Kobe, Hyōgo
  - Nishinomiya Municipal Central Hospital, Nishinomiya, Hyōgo
  - National Hospital Organization Kanazawa Medical Center, Kanazawa, Ishikawa-ken
  - Morita Hospital, Komatsu, Ishikawa-ken
  - Sagamidai Hospital, Zama, Kanagawa
  - Misugikai Medical Corporation Otokoyama Hospital, Yawata, Kyoto
  - National Hospital Organization Matsumoto Medical Center, Matsumoto, Nagano
  - Yodakubo Hospital, Nagawa-machi, Chisagata-gun, Nagano
  - National Hospital Organization Beppu Medical Center, Beppu, Oita Prefecture
  - National Hospital Organization Osaka Minami Medical Center, Kawachi-Nagano, Osaka
  - Kishiwada Tokushukai Hospital, Kishiwada, Osaka
  - Osaka Rosai Hospital, Sakai, Osaka
  - Nagayama Hospital, Sennan-gun, Osaka
  - Saiseikai Kawaguchi General Hospital, Kawaguchi, Saitama
  - Hanazono Orthopedics and Internal Medicine, Tokorozawa, Saitama
  - Japanese Red Cross Hamamatsu Hospital, Hamamatsu, Shizuoka
  - Iwata City Hospital, Iwata, Shizuoka
  - Tokyo Saiseikai Central Hospital, Minato-ku, Tokyo
  - Kitasato University Kitasato Institute Hospital, Minato-ku, Tokyo
  - National Hospital Organization Murayama Medical Center, Musashimurayama, Tokyo
  - Gate Town Hospital, Nerima-ku, Tokyo
  - Juntendo University Nerima Hospital, Nerima-ku, Tokyo
  - Nishikamata Orthopedic, Ōta-ku, Tokyo
  - AR-Ex Oyamadai Orthopedic, Setagaya-ku, Tokyo
  - Kohno Clinical Medicine Research Institute Daisan Kitashinagawa Hospital, Shinagawa-ku, Tokyo
  - Ohimachi Orthopaedic Clinic, Shinagawa-ku, Tokyo
  - Ogikubo Hospital, Suginami-ku, Tokyo
  - Medical Corporation Keiyukai Masumoto Orthopedic Clinic, Suginami-ku, Tokyo
  - Daido Hospital, Toshima-ku, Tokyo
  - Tonami General Hospital, Tonami, Toyama
  - Wakayama Medical University Kihoku Hospital, Ito-gun, Wakayama
  - Shimonoseki City Hospital, Shimonoseki-shi, Yamaguchi
  - Akita University Hospital, Akita
  - Kuroda Orthopedic Hospital, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - Morimoto Clinic, Osaka
  - Nagayoshi General Hospital, Osaka
  - Saitama Municipal Hospital, Saitama

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Konno SI, Nikaido T, Markman JD, Ohta M, Machida T, Isogawa N, Yoshimatsu H, Viktrup L, Brown MT, West CR, Verburg KM. Tanezumab for chronic low back pain: a long-term, randomized, celecoxib-controlled Japanese Phase III safety study. Pain Manag. 2022 Apr;12(3):323-335. doi: 10.2217/pmt-2021-0040. Epub 2021 Nov 17. PMID 34786956
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A4091063

RESULTS

PARTICIPANT FLOW:
Groups:
- Tanezumab 5 mg: Participants were randomized to receive tanezumab (PF-04383119) 5 milligram (mg) subcutaneous (SC) injection once every 8 weeks, from Day 1 up to Week 56 and oral placebo capsules matched to celecoxib, twice daily, from Day 1 up to Week 56. Participants were followed up for 24 weeks after last dose of study drug (maximum up to Week 80).
- Tanezumab 10 mg: Participants were randomized to receive tanezumab (PF-04383119) 10 mg SC injection once every 8 weeks, from Day 1 up to Week 56 and oral placebo capsules matched to celecoxib, twice daily, from Day 1 up to Week 56. Participants were followed up for 24 weeks after last dose of study drug (maximum up to Week 80).
- Celecoxib: Participants were randomized to receive celecoxib 100 mg capsules orally, twice daily, from Day 1 up to Week 56 and SC injection of placebo matched to tanezumab (PF-04383119) once every 8 weeks, from Day 1 up to Week 56. Participants were followed up for 24 weeks after last dose of study drug (maximum up to Week 80).
Period: Treatment Period (56 Weeks)
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Started | 92 | 93 | 92
Treated | 92 | 93 | 92
Completed | 62 | 43 | 43
Not Completed | 30 | 50 | 49
Not completed — Adverse Event | 3 | 5 | 4
Not completed — Lack of Efficacy | 1 | 4 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Other | 1 | 4 | 5
Not completed — Withdrawal by Subject | 0 | 1 | 4
Not completed — Not Met Protocol-Specified Criteria | 25 | 35 | 35
Period: Follow-up Period (24 Weeks)
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Started | 92 (All participants on either completion or discontinuation of treatment, entered follow up period.) | 93 (All participants on either completion or discontinuation of treatment, entered follow up period.) | 92 (All participants on either completion or discontinuation of treatment, entered follow up period.)
Completed | 88 | 82 | 87
Not Completed | 4 | 11 | 5
Not completed — Adverse Event | 1 | 1 | 0
Not completed — Lack of Efficacy | 0 | 2 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Other | 1 | 4 | 2
Not completed — Withdrawal by Subject | 1 | 3 | 3

BASELINE CHARACTERISTICS:
Population: Safety analysis population included all participants who were treated with tanezumab or placebo matched to tanezumab.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib | Total
Number analyzed (Participants) | 92 | 93 | 92 | 277
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.35 (12.97) | 52.32 (14.02) | 54.34 (14.21) | 53.33 (13.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 44 | 38 | 119
  Male | 55 | 49 | 54 | 158
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 92 | 93 | 92 | 277
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 92 | 93 | 92 | 277
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to 24 weeks after last dose of study drug (up to Week 80) that were absent before treatment or that worsened relative to pretreatment state. AEs included both serious and non-serious AEs.
Time Frame: Baseline (Day 1) up to 24 weeks after last dose of study drug (up to Week 80)
Population: Safety analysis population included all participants who were treated with tanezumab or placebo matched to tanezumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
Participants
  Participants with AEs | 70 | 63 | 67
  Participants with SAEs | 8 | 11 | 4

2. Primary Outcome: Number of Participants With Treatment-Emergent Treatment Related Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Treatment-related AE was any untoward medical occurrence attributed to study drug in participant who received study drug. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to 24 weeks after last dose of study drug (up to Week 80). Relatedness to study drug was assessed by the investigator. AEs included both serious and non-serious AEs.
Time Frame: Baseline up to 24 weeks after last dose of study drug (up to Week 80)
Population: Safety analysis population included all participants who were treated with tanezumab or placebo matched to tanezumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
Participants
  Participants with treatment related AEs | 11 | 7 | 12
  Participants with treatment related SAEs | 1 | 1 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Laboratory Test Abnormalities
Description: Abnormality criteria included: hemoglobin (HGB); hematocrit; erythrocytes < 0.8*lower limit of normal (LLN); erythrocyte mean corpuscular volume/HGB/ HGB concentration, erythrocytes distribution width <0.9*LLN, >1.1*upper limit of normal (ULN); platelets <0.5*LLN,>1.75* ULN; white blood cell count<0.6*LLN, >1.5*ULN; lymphocytes, leukocytes, neutrophils <0.8*LLN, >1.2*ULN; basophils, eosinophils, monocytes >1.2*ULN; total bilirubin>1.5*ULN; aspartate aminotransferase (AT), alanine AT, gamma glutamyl transferase, lactate dehydrogenase, alkaline phosphatase >3.0*ULN; total protein; albumin<0.8*LLN, >1.2*ULN; blood urea nitrogen, creatinine, cholesterol, triglycerides >1.3*ULN; urate >1.2*ULN; sodium <0.95*LLN,>1.05*ULN; potassium, chloride, calcium, magnesium, bicarbonate <0.9*LLN, >1.1*ULN; phosphate <0.8*LLN, >1.2*ULN; glucose <0.6*LLN, >1.5*ULN; HGB A1C >1.3*ULN; creatine kinase >2.0*ULN; nitrite >=1. Investigator judged clinical significance of laboratory test abnormalities.
Time Frame: Baseline up to Week 80
Population: Safety analysis population included all participants who were treated with tanezumab or placebo matched to tanezumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
Participants | 1 | 0 | 1

4. Primary Outcome: Number of Participants With Clinically Significant Vital Signs Abnormalities
Description: Vital signs included systolic blood pressure, diastolic blood pressure and pulse rate. Investigator judged clinical significance of vital signs' abnormalities.
Time Frame: Baseline up to Week 80
Population: Safety analysis population included all participants who were treated with tanezumab or placebo matched to tanezumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
Participants | 4 | 2 | 5

5. Primary Outcome: Number of Participants With Confirmed Orthostatic Hypotension From Baseline up to Week 80
Description: Orthostatic hypotension was defined as postural change (supine to standing) that met the following criteria: for systolic blood pressure (BP) less than or equal to (<=) 150 millimeter of mercury (mmHg) (mean supine): reduction in systolic BP >=20 mmHg or reduction in diastolic BP >=10 mmHg at the 1 and/or 3 minute standing BP measurements. For systolic BP greater than (>) 150 mmHg (mean supine): reduction in systolic BP >=30 mmHg or reduction in diastolic BP >=15 mmHg at the 1 and/or 3 minute standing BP measurements. If the 1 minute or 3 minute standing BP in a sequence met the orthostatic hypotension criteria, then that sequence was considered positive. If 2 of 2 or 2 of 3 sequences were positive, then orthostatic hypotension was considered confirmed.
Time Frame: Baseline up to Week 80
Population: Safety analysis population included all participants who were treated with tanezumab or placebo matched to tanezumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
Participants | 0 | 2 | 0

6. Primary Outcome: Change From Screening in Mean Total Symptom Impact Score as Per Survey of Autonomic Symptoms (SAS) at Week 24
Description: SAS is a participant rated 12 items questionnaire for males and 11 items questionnaire for females. SAS measures autonomic symptoms of neuropathy and their impact on participants' well-being, during the past 6 months. Each item was related to a symptom/health problem. At scheduled time points, participants were asked to answer "Yes" or "No" for each of symptoms/health problems experienced during past 6 months. If a participant answered "Yes" for a symptom, then impact of that symptom was rated on a 5 point scale, ranged from 1 (least sever impact) to 5 (most severe impact), where higher scores signified more severe impact of symptoms. The total symptom impact score was calculated as the sum of impact of all symptoms. Overall possible range for the total symptom impact score was 0 (no impact) to 60 (extreme impact) for males and 0 (no impact) to 55 (extreme impact) for females, higher scores indicated more severe impact of symptoms on participants' well-being.
Time Frame: Screening (up to 37 days before Day 1), Week 24
Population: Safety analysis population included all participants who were treated with tanezumab or placebo matched to tanezumab. Here, 'Number Analyzed' = participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
units on a scale
  Screening | 0.76 (1.51) | 0.86 (1.58) | 1.10 (1.78)
  Change at Week 24: number analyzed (Participants) | 63 | 46 | 46
  Change at Week 24 | 0.79 (2.29) | 0.93 (3.36) | 0.04 (2.66)

7. Primary Outcome: Change From Screening in Mean Total Symptom Impact Score as Per Survey of Autonomic Symptoms (SAS) at Week 56
Description: as for outcome 6
Time Frame: Screening, Week 56
Population: Safety analysis population included all participants who were treated with tanezumab or placebo matched to tanezumab. Here, "Overall number of participants analyzed" signifies only those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 62 | 43 | 43
units on a scale | 0.89 (3.30) | 0.86 (4.10) | 0.35 (2.60)

8. Primary Outcome: Change From Screening in Mean Total Symptom Impact Scores as Per Survey of Autonomic Symptoms (SAS) at Week 80
Description: as for outcome 6
Time Frame: Screening, Week 80
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 62 | 43 | 43
units on a scale | 0.69 (2.81) | 1.26 (3.29) | 0.72 (3.17)

9. Primary Outcome: Change From Screening in Mean Total Symptom Impact Score as Per Survey of Autonomic Symptoms (SAS) at Early Termination Follow-up Visit 1
Description: SAS: participant rated 12 items questionnaire for males; 11 items questionnaire for females. SAS measures autonomic symptoms of neuropathy and their impact on participants' well-being, during past 6 months. Each item was related to a symptom/health problem. At scheduled time points, participants answered "Yes" or "No" for each of symptoms/health problems experienced during past 6 months. If participant answered "Yes" for a symptom, then impact of that symptom was rated on 5 point scale (1 [least sever impact] to 5 [most severe impact]); higher scores = more severe impact of symptoms. Total impact score = sum of impact of all symptoms; range for males =0 (no impact) to 60 (extreme impact); females =0 (no impact) to 55 (extreme impact); higher scores = more severe impact of symptoms on participants' well-being. Participants discontinuing from study treatment before Week 56, had early termination follow-up visit 1 at 8 weeks after last dose of tanezumab or placebo matched to tanezumab.
Time Frame: Screening, Early Termination Follow-up Visit 1 (at 8 weeks after last dose of tanezumab or placebo matched to tanezumab)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 30 | 49 | 48
units on a scale | 2.50 (5.28) | 0.82 (3.42) | 2.15 (3.94)

10. Primary Outcome: Change From Screening in Mean Total Symptom Impact Scores as Per Survey of Autonomic Symptoms (SAS) at Early Termination Follow-up Visit 3
Description: SAS: participant rated 12 items questionnaire for males; 11 items questionnaire for females. SAS measures autonomic symptoms of neuropathy and their impact on participants' well-being, during past 6 months. Each item was related to a symptom/health problem. At scheduled time points, participants answered "Yes" or "No" for each of symptoms/health problems experienced during past 6 months. If participant answered "Yes" for a symptom, then impact of that symptom was rated on 5 point scale (1 [least sever impact] to 5 [most severe impact]); higher scores = more severe impact of symptoms. Total impact score = sum of impact of all symptoms; range for males =0 (no impact) to 60 (extreme impact); females =0 (no impact) to 55 (extreme impact); higher scores = more severe impact of symptoms on participants' well-being. Participants discontinuing from study treatment before Week 56, had early termination follow-up visit 3 at 24 weeks after last dose of tanezumab or placebo matched to tanezumab.
Time Frame: Screening, Early Termination Follow-up Visit 3 (at 24 weeks after last dose of tanezumab or placebo matched to tanezumab)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 27 | 45 | 43
units on a scale | 1.89 (5.57) | 1.60 (3.82) | 0.88 (3.03)

11. Primary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Assessments
Description: Electrocardiogram assessment included PR, QRS, QT, QT interval corrected using Fridericia's formula (QTcF), QT interval corrected using Bazett's formula (QTcB), RR intervals, and heart rate. Investigator judged clinical significance of electrocardiogram assessment.
Time Frame: Baseline up to Week 16
Population: Safety analysis population included all participants who were treated with tanezumab or placebo matched to tanezumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
Participants | 2 | 0 | 2

12. Primary Outcome: Percentage of Participants With Individual Adjudicated Joint Safety Outcome/Event
Description: Percentage of participants with individual joint safety adjudication outcomes: rapidly progressive osteoarthritis (OA) type-1 only, rapidly progressive OA type-2 only, primary osteonecrosis, pathological fracture and subchondral insufficiency fracture is reported. Rapidly progressive (RP) OA type 1 events were those that the adjudication committee considered to have significant loss of joint space width >= 2 millimeter within approximately 1 year without gross structural failure. RP OA type 2 events were those considered to have destruction of bone including limited or total collapse of at least 1 subchondral surface that is not normally present in conventional end-stage osteoarthritis. Subchondral insufficiency fractures are a type of stress fractures which occur below the cartilage on the weight bearing surface of a bone.
Time Frame: Baseline up to Week 80
Population: Safety analysis population included all participants who were treated with tanezumab or placebo matched to tanezumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
percentage of participants
  Rapidly Progressive OA type 1 | 1 [0.0 to 5.9] | 0 [0.0 to 3.9] | 0 [0.0 to 3.9]
  Rapidly Progressive OA type 2 | 0 [0.0 to 3.9] | 1 [0.0 to 5.8] | 0 [0.0 to 3.9]
  Primary Osteonecrosis | 0 [0.0 to 3.9] | 0 [0.0 to 3.9] | 0 [0.0 to 3.9]
  Pathological Fracture | 0 [0.0 to 3.9] | 0 [0.0 to 3.9] | 0 [0.0 to 3.9]
  Subchondral Insufficiency Fracture | 0 [0.0 to 3.9] | 1 [0.0 to 5.8] | 0 [0.0 to 3.9]

13. Primary Outcome: Observation Time-Adjusted Event Rate for an Individual Adjudicated Joint Safety Outcome/Event
Description: Individual adjudicated joint safety outcomes/event: rapidly progressive OA (type-1,type-2), primary osteonecrosis, pathological fracture and subchondral insufficiency fracture. Observation time was defined as the start day of first SC study medication until either the (i) date of completion of or withdrawal from study, if a participant did not have the event, or (ii) date of the event (earliest event within each participant in the case of multiple events). Event rate for any individual adjudicated joint safety outcome/event = the number of events per 1000 participant-years at risk.
Time Frame: Baseline (Day 1) up to Week 80
Population: Safety analysis population included all participants who were treated with tanezumab or placebo matched to tanezumab.
Measure: Number (95% Confidence Interval); unit: events per 1000 participant-years
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
events per 1000 participant-years
  Rapidly Progressive OA Type 1 | 8.9 [1.2 to 62.9] | 0 [0 to 0] | 0 [0 to 0]
  Rapidly Progressive OA Type 2 | 0 [0 to 0] | 10.4 [1.5 to 74.1] | 0 [0 to 0]
  Primary Osteonecrosis | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Pathological Fracture | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Subchondral Insufficiency Fracture | 0 [0 to 0] | 10.5 [1.5 to 74.6] | 0 [0 to 0]

14. Primary Outcome: Percentage of Participants With At Least 1 Total Joint Replacement
Description: Percentage of participants with at least 1 total knee, total hip or total shoulder joint replacement were reported.
Time Frame: Baseline (Day 1) up to Week 80
Population: Safety analysis population included all participants who were treated with tanezumab or placebo matched to tanezumab.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
percentage of participants | 0 [0.0 to 3.9] | 1 [0.0 to 5.8] | 0 [0.0 to 3.9]

15. Primary Outcome: Observation Time-Adjusted Event Rate for Total Joint Replacement (TJR) Event
Description: Observation time was defined as the start day of first SC study medication until either the (i) date of completion of or withdrawal from study, if a participant had no TJR, or (ii) date of TJR (earliest TJR within each participant in the case of multiple TJRs). Event rate = number of events per 1000 participant-years at risk.
Time Frame: Baseline (Day 1) up to Week 80
Population: Safety analysis population included all participants who were treated with tanezumab or placebo matched to tanezumab.
Measure: Number (95% Confidence Interval); unit: events per 1000 participant-years
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
events per 1000 participant-years | 0 [0 to 0] | 10.4 [1.5 to 74.1] | 0 [0 to 0]

16. Primary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Week 2
Description: NIS is a standardized instrument used to evaluate signs of peripheral neuropathy in participants. NIS is the sum of scores of 37 items, from both the left and right side of following 4 domains: cranial nerves (5 items), muscle weakness (19 items), reflexes (5 items) and sensation (8 items). Each of 24 items related to cranial nerves and muscle weakness, scored from 0 (normal) to 4 (paralysis); higher scores indicated higher abnormality/impairment. Each of 13 items related to reflexes and sensation, scored as 0 (normal), 1 (decreased) and 2 (absent); higher scores indicated lesser reflexes and sensation. For NIS possible overall score (combined of both left and right sides of each domain), ranged from 0 (no impairment) to 244 (maximum impairment), higher scores indicated increased/more neuropathic deficits.
Time Frame: Baseline, Week 2
Population: Safety analysis population included all participants who were treated with tanezumab or placebo matched to tanezumab.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
units on a scale
  Baseline | 0.84 (2.39) | 1.01 (4.06) | 0.87 (2.19)
  Change at Week 2 | -0.04 (0.25) | -0.01 (0.48) | 0.11 (1.19)

17. Primary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Week 4
Description: as for outcome 16
Time Frame: Baseline, Week 4
Population: Safety analysis population included all participants who were treated with tanezumab or placebo matched to tanezumab.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
units on a scale | -0.08 (0.50) | -0.02 (0.68) | 0.11 (1.08)

18. Primary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Week 8
Description: as for outcome 16
Time Frame: Baseline, Week 8
Population: Safety analysis population included all participants who were treated with tanezumab or placebo matched to tanezumab.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
units on a scale | -0.04 (0.39) | 0.15 (0.78) | 0.13 (0.99)

19. Primary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Week 16
Description: as for outcome 16
Time Frame: Baseline, Week 16
Population: Safety analysis population included all participants who were treated with tanezumab or placebo matched to tanezumab.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
units on a scale | -0.02 (0.21) | 0.05 (0.71) | 0.01 (0.87)

20. Primary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Week 24
Description: as for outcome 16
Time Frame: Baseline, Week 24
Population: Safety analysis population included all participants who were treated with tanezumab or placebo matched to tanezumab.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
units on a scale | -0.02 (0.21) | 0.09 (0.70) | 0.28 (1.83)

21. Primary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Week 32
Description: as for outcome 16
Time Frame: Baseline, Week 32
Population: Safety analysis population included all participants who were treated with tanezumab or placebo matched to tanezumab.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
units on a scale | 0.00 (0.36) | -0.01 (0.96) | 0.04 (1.64)

22. Primary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Week 40
Description: as for outcome 16
Time Frame: Baseline, Week 40
Population: Safety analysis population included all participants who were treated with tanezumab or placebo matched to tanezumab.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
units on a scale | 0.14 (1.14) | 0.04 (1.03) | 0.04 (1.64)

23. Primary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Week 48
Description: as for outcome 16
Time Frame: Baseline, Week 48
Population: Safety analysis population included all participants who were treated with tanezumab or placebo matched to tanezumab.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
units on a scale | 0.09 (1.09) | -0.01 (0.97) | 0.04 (1.70)

24. Primary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Week 56
Description: as for outcome 16
Time Frame: Baseline, Week 56
Population: Safety analysis population included all participants who were treated with tanezumab or placebo matched to tanezumab.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
units on a scale | 0.09 (1.09) | -0.02 (0.97) | 0.04 (1.64)

25. Primary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Week 64
Description: as for outcome 16
Time Frame: Baseline, Week 64
Population: Safety analysis population included all participants who were treated with tanezumab or placebo matched to tanezumab.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
units on a scale | 0.18 (1.43) | 0.01 (0.98) | 0.04 (1.70)

26. Primary Outcome: Change From Baseline in Neuropathy Impairment Score (NIS) at Week 80
Description: as for outcome 16
Time Frame: Baseline, Week 80
Population: Safety analysis population included all participants who were treated with tanezumab or placebo matched to tanezumab.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
units on a scale | 0.03 (1.26) | 0.00 (0.97) | 0.17 (2.36)

27. Primary Outcome: Largest Change From Baseline in Neuropathy Impairment Score (NIS) to Any Post-baseline Visit
Description: NIS is a standardized instrument used to evaluate signs of peripheral neuropathy in participants. NIS is the sum of scores of 37 items, from both the left and right side of following 4 domains: cranial nerves (5 items), muscle weakness (19 items), reflexes (5 items) and sensation (8 items). Each of 24 items related to cranial nerves and muscle weakness, scored from 0 (normal) to 4 (paralysis); higher scores indicated higher abnormality/impairment. Each of 13 items related to reflexes and sensation, scored as 0 (normal), 1 (decreased) and 2 (absent); higher scores indicated lesser reflexes and sensation. For NIS possible overall score (combined of both left and right sides of each domain), ranged from 0 (no impairment) to 244 (maximum impairment), higher scores indicated increased/more neuropathic deficits. Largest change from baseline here means worst post- baseline change value (among all change from baseline values).
Time Frame: Baseline to any post-baseline visit (until Week 80)
Population: Safety analysis population included all participants who were treated with tanezumab or placebo matched to tanezumab.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
units on a scale | 0.33 (1.47) | 0.37 (1.06) | 0.78 (2.62)

28. Primary Outcome: Number of Participants With Anti Tanezumab Antibodies From Baseline up to Week 80
Description: Human serum samples were analyzed for the presence or absence of anti-tanezumab antibodies by using a validated analytical method. Number of participants with presence of anti-tanezumab antibodies are reported.
Time Frame: Baseline up to Week 80
Population: Safety analysis population included all participants who were treated with tanezumab or placebo matched to tanezumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
Participants | 21 | 41 | 62

29. Secondary Outcome: Change From Baseline in Average Low Back Pain Intensity (LBPI) at Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48, and 56: Multiple Imputation
Description: Average LBPI was assessed on an 11-point numeric rating scale (NRS). Participants described their average LBPI during the past 24 hours (at each specified/scheduled time-point) on a scale ranging from 0 (no pain) to 10 (worst possible pain), where higher scores indicated worse pain.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48 and 56
Population: Intent to treat (ITT) population included all randomized participants who received at least 1 dose of SC study medication (either tanezumab or placebo matched to tanezumab). Missing data were imputed with multiple imputation method based on the reason for missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
units on a scale
  Change at Week 2 | -0.47 (0.14) | -0.69 (0.14) | -0.46 (0.14)
  Change at Week 4 | -0.83 (0.17) | -1.05 (0.17) | -0.56 (0.17)
  Change at Week 8 | -1.24 (0.20) | -1.64 (0.20) | -1.07 (0.20)
  Change at Week 12 | -2.19 (0.23) | -2.46 (0.23) | -1.85 (0.23)
  Change at Week 16 | -2.91 (0.23) | -2.51 (0.23) | -2.28 (0.23)
  Change at Week 24 | -2.88 (0.28) | -2.41 (0.28) | -2.11 (0.29)
  Change at Week 32 | -2.95 (0.29) | -2.34 (0.30) | -2.08 (0.30)
  Change at Week 40 | -3.00 (0.30) | -2.32 (0.30) | -2.06 (0.29)
  Change at Week 48 | -3.07 (0.30) | -2.31 (0.31) | -2.09 (0.31)
  Change at Week 56 | -2.98 (0.29) | -2.22 (0.30) | -2.13 (0.30)
Statistical Analysis 1: Comparison: Tanezumab 5 mg vs Celecoxib; Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as a fixed effect, and baseline average LBPI as a covariates, and study site as a random effect; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.01, 95% CI 2-sided [-0.38 to 0.35], Standard Error of Mean 0.18
Statistical Analysis 2: Comparison: Tanezumab 10 mg vs Celecoxib; [analysis description as in outcome 29, analysis 1]; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.24, 95% CI 2-sided [-0.60 to 0.13], Standard Error of Mean 0.19
Statistical Analysis 3: Comparison: Tanezumab 5 mg vs Celecoxib; Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as a fixed effect, and baseline average LBPI as a covariates, and study site as a random effect; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.27, 95% CI 2-sided [-0.70 to 0.15], Standard Error of Mean 0.22
Statistical Analysis 4: Comparison: Tanezumab 10 mg vs Celecoxib; [analysis description as in outcome 29, analysis 3]; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.50, 95% CI 2-sided [-0.93 to -0.07], Standard Error of Mean 0.22
Statistical Analysis 5: Comparison: Tanezumab 5 mg vs Celecoxib; Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as a fixed effect, and baseline average LBPI as a covariates, and study site as a random effect; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.18, 95% CI 2-sided [-0.69 to 0.33], Standard Error of Mean 0.26
Statistical Analysis 6: Comparison: Tanezumab 10 mg vs Celecoxib; [analysis description as in outcome 29, analysis 5]; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.57, 95% CI 2-sided [-1.09 to -0.06], Standard Error of Mean 0.26
Statistical Analysis 7: Comparison: Tanezumab 5 mg vs Celecoxib; Week 12: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as a fixed effect, and baseline average LBPI as a covariates, and study site as a random effect; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.34, 95% CI 2-sided [-0.94 to 0.27], Standard Error of Mean 0.31
Statistical Analysis 8: Comparison: Tanezumab 10 mg vs Celecoxib; [analysis description as in outcome 29, analysis 7]; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.60, 95% CI 2-sided [-1.21 to 0.00], Standard Error of Mean 0.31
Statistical Analysis 9: Comparison: Tanezumab 5 mg vs Celecoxib; Week 16: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as a fixed effect, and baseline average LBPI as a covariates, and study site as a random effect; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.63, 95% CI 2-sided [-1.24 to -0.03], Standard Error of Mean 0.31
Statistical Analysis 10: Comparison: Tanezumab 10 mg vs Celecoxib; [analysis description as in outcome 29, analysis 9]; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.23, 95% CI 2-sided [-0.84 to 0.38], Standard Error of Mean 0.31
Statistical Analysis 11: Comparison: Tanezumab 5 mg vs Celecoxib; Week 24: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as a fixed effect, and baseline average LBPI as a covariates, and study site as a random effect; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.76, 95% CI 2-sided [-1.53 to 0.01], Standard Error of Mean 0.39
Statistical Analysis 12: Comparison: Tanezumab 10 mg vs Celecoxib; [analysis description as in outcome 29, analysis 11]; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.30, 95% CI 2-sided [-1.07 to 0.47], Standard Error of Mean 0.39
Statistical Analysis 13: Comparison: Tanezumab 5 mg vs Celecoxib; Week 32: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as a fixed effect, and baseline average LBPI as a covariates, and study site as a random effect; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.87, 95% CI 2-sided [-1.65 to -0.08], Standard Error of Mean 0.40
Statistical Analysis 14: Comparison: Tanezumab 10 mg vs Celecoxib; [analysis description as in outcome 29, analysis 13]; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.25, 95% CI 2-sided [-1.06 to 0.55], Standard Error of Mean 0.41
Statistical Analysis 15: Comparison: Tanezumab 5 mg vs Celecoxib; Week 40: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as a fixed effect, and baseline average LBPI as a covariates, and study site as a random effect; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.94, 95% CI 2-sided [-1.72 to -0.15], Standard Error of Mean 0.40
Statistical Analysis 16: Comparison: Tanezumab 10 mg vs Celecoxib; [analysis description as in outcome 29, analysis 15]; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.26, 95% CI 2-sided [-1.05 to 0.54], Standard Error of Mean 0.41
Statistical Analysis 17: Comparison: Tanezumab 5 mg vs Celecoxib; Week 48: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as a fixed effect, and baseline average LBPI as a covariates, and study site as a random effect; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.97, 95% CI 2-sided [-1.80 to -0.15], Standard Error of Mean 0.42
Statistical Analysis 18: Comparison: Tanezumab 10 mg vs Celecoxib; [analysis description as in outcome 29, analysis 17]; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.22, 95% CI 2-sided [-1.04 to 0.61], Standard Error of Mean 0.42
Statistical Analysis 19: Comparison: Tanezumab 5 mg vs Celecoxib; Week 56: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as a fixed effect, and baseline average LBPI as a covariates, and study site as a random effect; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.85, 95% CI 2-sided [-1.65 to -0.05], Standard Error of Mean 0.41
Statistical Analysis 20: Comparison: Tanezumab 10 mg vs Celecoxib; [analysis description as in outcome 29, analysis 19]; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.09, 95% CI 2-sided [-0.88 to 0.71], Standard Error of Mean 0.41

30. Secondary Outcome: Change From Baseline in Average Low Back Pain Intensity (LBPI) at Week 64: Observed Data
Description: Average LBPI was assessed on an 11-point NRS. Participants described their average LBPI during the past 24 hours (at each specified/scheduled time-point) on a scale ranging from 0 (no pain) to 10 (worst possible pain), where higher scores indicated worse pain.
Time Frame: Baseline, Week 64
Population: ITT population analyzed. ''Overall number of participants analyzed'' = participants who were evaluable for this outcome measure. Observed data: analysis was performed using all available data at Week 64, and no imputation technique was used for missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 61 | 43 | 43
units on a scale | -3.60 (1.81) | -3.96 (1.82) | -3.46 (1.89)

31. Secondary Outcome: Change From Baseline in Roland-Morris Disability Questionnaire (RMDQ) Total Scores at Weeks 2, 4, 8, 16, 24, 32, 40, 48, and 56: Multiple Imputation
Description: The RMDQ is a self-administered, widely used health status measure index of how well participants with low back pain (LBP) are able to function with regard to daily activities. It measures pain and function, using 24 items describing limitations to everyday life that can be caused by LBP. Participants were asked to check/select only those items out of 24 items, which described them at each specified time point. The total number of items checked in questionnaire was equal to RMDQ total score, overall possible score ranging from 0 (no disability) to 24 (maximum disability), where higher scores indicated greater/more disability.
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 32, 40, 48 and 56
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or placebo matched to tanezumab). Missing data were imputed with multiple imputation method based on the reason for missing data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
units on a scale
  Change at Week 2 | -2.09 (0.34) | -2.09 (0.34) | -1.23 (0.34)
  Change at Week 4 | -2.41 (0.40) | -2.35 (0.40) | -1.89 (0.39)
  Change at Week 8 | -2.74 (0.39) | -3.23 (0.39) | -2.68 (0.39)
  Change at Week 16 | -3.85 (0.41) | -4.38 (0.42) | -3.84 (0.42)
  Change at Week 24 | -3.58 (0.48) | -3.32 (0.47) | -3.16 (0.48)
  Change at Week 32 | -3.62 (0.48) | -3.11 (0.49) | -3.02 (0.49)
  Change at Week 40 | -3.98 (0.50) | -2.95 (0.50) | -2.90 (0.51)
  Change at Week 48 | -3.99 (0.48) | -2.96 (0.51) | -3.19 (0.50)
  Change at Week 56 | -3.95 (0.49) | -2.91 (0.50) | -2.94 (0.50)
Statistical Analysis 1: Comparison: Tanezumab 5 mg vs Celecoxib; Week 2: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline RMDQ as covariates, and study site as a random effect; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.86, 95% CI 2-sided [-1.77 to 0.04], Standard Error of Mean 0.46
Statistical Analysis 2: Comparison: Tanezumab 10 mg vs Celecoxib; [analysis description as in outcome 31, analysis 1]; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -1.05, 95% CI 2-sided [-1.96 to -0.14], Standard Error of Mean 0.46
Statistical Analysis 3: Comparison: Tanezumab 5 mg vs Celecoxib; Week 4: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline RMDQ as covariates, and study site as a random effect; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.52, 95% CI 2-sided [-1.48 to 0.43], Standard Error of Mean 0.49
Statistical Analysis 4: Comparison: Tanezumab 10 mg vs Celecoxib; [analysis description as in outcome 31, analysis 3]; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.46, 95% CI 2-sided [-1.43 to 0.51], Standard Error of Mean 0.50
Statistical Analysis 5: Comparison: Tanezumab 5 mg vs Celecoxib; Week 8: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline RMDQ as covariates, and study site as a random effect; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.06, 95% CI 2-sided [-1.04 to 0.91], Standard Error of Mean 0.50
Statistical Analysis 6: Comparison: Tanezumab 10 mg vs Celecoxib; [analysis description as in outcome 31, analysis 5]; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.55, 95% CI 2-sided [-1.53 to 0.44], Standard Error of Mean 0.50
Statistical Analysis 7: Comparison: Tanezumab 5 mg vs Celecoxib; Week 16: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline RMDQ as covariates, and study site as a random effect; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.01, 95% CI 2-sided [-1.06 to 1.05], Standard Error of Mean 0.54
Statistical Analysis 8: Comparison: Tanezumab 10 mg vs Celecoxib; [analysis description as in outcome 31, analysis 7]; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.53, 95% CI 2-sided [-1.60 to 0.53], Standard Error of Mean 0.54
Statistical Analysis 9: Comparison: Tanezumab 5 mg vs Celecoxib; Week 24: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline RMDQ as covariates, and study site as a random effect; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.42, 95% CI 2-sided [-1.71 to 0.88], Standard Error of Mean 0.66
Statistical Analysis 10: Comparison: Tanezumab 10 mg vs Celecoxib; [analysis description as in outcome 31, analysis 9]; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.16, 95% CI 2-sided [-1.47 to 1.14], Standard Error of Mean 0.66
Statistical Analysis 11: Comparison: Tanezumab 5 mg vs Celecoxib; Week 32: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline RMDQ as covariates, and study site as a random effect; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.60, 95% CI 2-sided [-1.90 to 0.71], Standard Error of Mean 0.67
Statistical Analysis 12: Comparison: Tanezumab 10 mg vs Celecoxib; [analysis description as in outcome 31, analysis 11]; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.09, 95% CI 2-sided [-1.44 to 1.25], Standard Error of Mean 0.69
Statistical Analysis 13: Comparison: Tanezumab 5 mg vs Celecoxib; Week 40: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline RMDQ as covariates, and study site as a random effect; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -1.08, 95% CI 2-sided [-2.43 to 0.28], Standard Error of Mean 0.69
Statistical Analysis 14: Comparison: Tanezumab 10 mg vs Celecoxib; [analysis description as in outcome 31, analysis 13]; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.04, 95% CI 2-sided [-1.41 to 1.32], Standard Error of Mean 0.70
Statistical Analysis 15: Comparison: Tanezumab 5 mg vs Celecoxib; Week 48: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline RMDQ as covariates, and study site as a random effect; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -0.80, 95% CI 2-sided [-2.17 to 0.57], Standard Error of Mean 0.70
Statistical Analysis 16: Comparison: Tanezumab 10 mg vs Celecoxib; [analysis description as in outcome 31, analysis 15]; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = 0.24, 95% CI 2-sided [-1.16 to 1.64], Standard Error of Mean 0.71
Statistical Analysis 17: Comparison: Tanezumab 5 mg vs Celecoxib; Week 56: Multiple imputation method was applied for missing data, with imputation dependent on reason for missing data. ANCOVA model for imputed datasets included treatment as fixed effects, baseline RMDQ as covariates, and study site as a random effect; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = -1.01, 95% CI 2-sided [-2.37 to 0.35], Standard Error of Mean 0.69
Statistical Analysis 18: Comparison: Tanezumab 10 mg vs Celecoxib; [analysis description as in outcome 31, analysis 17]; Test type: Other — No formal hypotheses were tested in the study; LS Mean Difference = 0.03, 95% CI 2-sided [-1.35 to 1.42], Standard Error of Mean 0.71

32. Secondary Outcome: Change From Baseline in Roland-Morris Disability Questionnaire (RMDQ) Total Score at Week 64: Observed Data
Description: as for outcome 31
Time Frame: Baseline, Week 64
Population: ITT population analyzed. "Overall number of participants analyzed" = participants who were evaluable for this outcome measure. Observed data: analysis was performed using all available data at Week 64 and no imputation technique was used for missing data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 62 | 43 | 43
units on a scale | -4.55 (4.04) | -5.72 (4.61) | -5.02 (3.96)

33. Secondary Outcome: Change From Baseline in the Patient's Global Assessment (PGA) of Low Back Pain at Weeks 2, 4, 8, 16, 24, 32, 40, 48, 56 and 64
Description: PGA of low back pain was assessed by asking a question to participants: "Considering all the ways your low back pain affects you, how are you doing today?" Participants responded on a 5 point Likert scale ranging from 1 to 5, using interactive response technology (IRT), where 1= very good (asymptomatic and no limitation of normal activities); 2= good (mild symptoms and no limitation of normal activities); 3= fair (moderate symptoms and limitation of some normal activities); 4= poor (severe symptoms and inability to carry out most normal activities); and 5= very poor (very severe symptoms which are intolerable and inability to carry out all normal activities). Higher scores indicated worsening of condition.
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 32, 40, 48, 56 and 64
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or placebo matched to tanezumab). Here, 'Number Analyzed' = participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
units on a scale
  Baseline | 3.24 (0.45) | 3.14 (0.38) | 3.13 (0.34)
  Change at Week 2 | -0.43 (0.63) | -0.40 (0.63) | -0.28 (0.52)
  Change at Week 4: number analyzed (Participants) | 92 | 92 | 91
  Change at Week 4 | -0.48 (0.72) | -0.46 (0.73) | -0.37 (0.59)
  Change at Week 8: number analyzed (Participants) | 92 | 92 | 90
  Change at Week 8 | -0.62 (0.74) | -0.66 (0.77) | -0.44 (0.66)
  Change at Week 16: number analyzed (Participants) | 91 | 89 | 88
  Change at Week 16 | -0.92 (0.75) | -0.82 (0.72) | -0.81 (0.74)
  Change at Week 24: number analyzed (Participants) | 63 | 50 | 48
  Change at Week 24 | -1.10 (0.69) | -1.22 (0.62) | -0.96 (0.62)
  Change at Week 32: number analyzed (Participants) | 63 | 46 | 46
  Change at Week 32 | -1.14 (0.69) | -1.13 (0.65) | -0.91 (0.55)
  Change at Week 40: number analyzed (Participants) | 63 | 45 | 44
  Change at Week 40 | -1.29 (0.73) | -1.09 (0.60) | -1.02 (0.59)
  Change at Week 48: number analyzed (Participants) | 63 | 45 | 44
  Change at Week 48 | -1.21 (0.70) | -1.11 (0.57) | -1.02 (0.66)
  Change at Week 56: number analyzed (Participants) | 63 | 43 | 43
  Change at Week 56 | -1.13 (0.68) | -1.14 (0.56) | -1.07 (0.59)
  Change at Week 64: number analyzed (Participants) | 62 | 43 | 43
  Change at Week 64 | -0.94 (0.72) | -0.84 (0.61) | -0.86 (0.71)

34. Secondary Outcome: Percentage of Participants With Cumulative Percent Change From Baseline in Average Low Back Pain Intensity (LBPI) Score at Weeks 16, 24 and 56
Description: Average LBPI was assessed on an 11-point numeric rating scale (NRS). Participants described their average LBPI during the past 24 hours (at each specified/scheduled time point) on a scale ranging from 0 (no pain) to 10 (worst possible pain), where higher scores indicated worse pain. Percentage of participants with cumulative reduction (as percent change) (greater than [>] 0%; >= 10, 20, 30, 40, 50, 60, 70, 80, 90 and equals to [=] 100%) in average LBPI from baseline to weeks 16, 24 and 56 were reported. Participants (%) might have been counted more than once under various rows.
Time Frame: Baseline, Weeks 16, 24 and 56
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or placebo matched to tanezumab).
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
percentage of participants
  Week 16: >0% | 89.1 | 81.7 | 81.5
  Week 16: >=10% | 85.9 | 77.4 | 78.3
  Week 16: >=20% | 76.1 | 67.7 | 66.3
  Week 16: >=30% | 71.7 | 57.0 | 58.7
  Week 16: >=40% | 59.8 | 46.2 | 45.7
  Week 16: >=50% | 51.1 | 35.5 | 32.6
  Week 16: >=60% | 33.7 | 25.8 | 16.3
  Week 16: >=70% | 19.6 | 17.2 | 8.7
  Week 16: >=80% | 13.0 | 14.0 | 6.5
  Week 16: >=90% | 3.3 | 4.3 | 2.2
  Week 16: =100% | 3.3 | 4.3 | 2.2
  Week 24: >0% | 72.8 | 60.2 | 59.8
  Week 24: >=10% | 70.7 | 57.0 | 57.6
  Week 24: >=20% | 69.6 | 55.9 | 55.4
  Week 24: >=30% | 65.2 | 51.6 | 53.3
  Week 24: >=40% | 57.6 | 48.4 | 46.7
  Week 24: >=50% | 50.0 | 43.0 | 38.0
  Week 24: >=60% | 38.0 | 35.5 | 20.7
  Week 24: >=70% | 25.0 | 21.5 | 10.9
  Week 24: >=80% | 17.4 | 16.1 | 4.3
  Week 24: >=90% | 6.5 | 4.3 | 1.1
  Week 24: =100% | 2.2 | 3.2 | 0
  Week 56: >=0% | 68.5 | 51.6 | 52.2
  Week 56: >=10% | 68.5 | 50.5 | 51.1
  Week 56: >=20% | 64.1 | 50.5 | 51.1
  Week 56: >=30% | 63.0 | 47.3 | 51.1
  Week 56: >=40% | 59.8 | 43.0 | 44.6
  Week 56: >=50% | 53.3 | 38.7 | 41.3
  Week 56: >=60% | 41.3 | 33.3 | 32.6
  Week 56: >=70% | 35.9 | 25.8 | 17.4
  Week 56: >=80% | 23.9 | 14.0 | 10.9
  Week 56: >=90% | 9.8 | 4.3 | 1.1
  Week 56: =100% | 4.3 | 2.2 | 1.1

35. Secondary Outcome: Percentage of Participants With >=30 Percent (%), >=50%, >=70% and >=90% Reduction From Baseline in Weekly Average Low Back Pain Intensity (LBPI) Score at Weeks 16, 24, 40 and 56
Description: Average LBPI was assessed on an 11-point numeric rating scale (NRS). Participants described their average LBPI during the past 24 hours (at each specified/scheduled time point) on a scale ranging from 0 (no pain) to 10 (worst possible pain), where higher scores indicated worse pain. Percentage of participants with reduction in average LBPI of at least (>=) 30%, 50%, 70% and 90% at Weeks 16, 24, 40, and 56 compared to baseline are reported here. Participants (%) might have been counted more than once under various rows.
Time Frame: Baseline, Weeks 16, 24, 40 and 56
Population: as for outcome 34
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
percentage of participants
  Week 16: At least 30% reduction | 71.7 [61.8 to 80.0] | 57.0 [46.8 to 66.6] | 58.7 [48.5 to 68.2]
  Week 16: At least 50% reduction | 51.1 [41.0 to 61.1] | 35.5 [26.5 to 45.6] | 32.6 [23.9 to 42.7]
  Week 16: At least 70% reduction | 19.6 [12.7 to 28.9] | 17.2 [10.8 to 26.2] | 8.7 [4.3 to 16.4]
  Week 16: At least 90% reduction | 3.3 [0.7 to 9.6] | 4.3 [1.3 to 10.9] | 2.2 [0.1 to 8.1]
  Week 24: At least 30% reduction | 65.2 [55.0 to 74.2] | 51.6 [41.6 to 61.5] | 53.3 [43.1 to 63.1]
  Week 24: At least 50% reduction | 50.0 [40.0 to 60.0] | 43.0 [33.4 to 53.2] | 38.0 [28.8 to 48.3]
  Week 24: At least 70% reduction | 25.0 [17.2 to 34.8] | 21.5 [14.3 to 31.0] | 10.9 [5.8 to 19.0]
  Week 24: At least 90% reduction | 6.5 [2.8 to 13.8] | 4.3 [1.3 to 10.9] | 1.1 [0.0 to 6.5]
  Week 40: At least 30% reduction | 66.3 [56.1 to 75.2] | 48.4 [38.5 to 58.4] | 48.9 [38.9 to 59.0]
  Week 40: At least 50% reduction | 53.3 [43.1 to 63.1] | 40.9 [31.4 to 51.0] | 35.9 [26.8 to 46.1]
  Week 40: At least 70% reduction | 34.8 [25.8 to 45.0] | 24.7 [17.0 to 34.4] | 17.4 [10.9 to 26.5]
  Week 40: At least 90% reduction | 7.6 [3.5 to 15.1] | 5.4 [2.0 to 12.3] | 0 [0.0 to 4.8]
  Week 56: At least 30% reduction | 63.0 [52.8 to 72.2] | 47.3 [37.5 to 57.4] | 51.1 [41.0 to 61.1]
  Week 56: At least 50% reduction | 53.3 [43.1 to 63.1] | 38.7 [29.4 to 48.9] | 41.3 [31.8 to 51.5]
  Week 56: At least 70% reduction | 35.9 [26.8 to 46.1] | 25.8 [17.9 to 35.6] | 17.4 [10.9 to 26.5]
  Week 56: At least 90% reduction | 9.8 [5.0 to 17.8] | 4.3 [1.3 to 10.9] | 1.1 [0.0 to 6.5]
Statistical Analysis 1: Comparison: Tanezumab 5 mg vs Celecoxib; Week 16: >=30%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = 13.0, 95% CI 2-sided [-0.8 to 26.3]
Statistical Analysis 2: Comparison: Tanezumab 10 mg vs Celecoxib; Week 16: >=30%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = -1.7, 95% CI 2-sided [-15.8 to 12.4]
Statistical Analysis 3: Comparison: Tanezumab 5 mg vs Celecoxib; Week 16: >=50%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = 18.5, 95% CI 2-sided [4.2 to 32.0]
Statistical Analysis 4: Comparison: Tanezumab 10 mg vs Celecoxib; Week 16: >=50%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = 2.9, 95% CI 2-sided [-10.7 to 16.3]
Statistical Analysis 5: Comparison: Tanezumab 5 mg vs Celecoxib; Week 16: >=70%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = 10.9, 95% CI 2-sided [0.6 to 20.7]
Statistical Analysis 6: Comparison: Tanezumab 10 mg vs Celecoxib; Week 16: >=70%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = 8.5, 95% CI 2-sided [-1.4 to 18.1]
Statistical Analysis 7: Comparison: Tanezumab 5 mg vs Celecoxib; Week 16: >=90%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = 1.1, 95% CI 2-sided [-4.3 to 6.5]
Statistical Analysis 8: Comparison: Tanezumab 10 mg vs Celecoxib; Week 16: >=90%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = 2.1, 95% CI 2-sided [-3.7 to 7.8]
Statistical Analysis 9: Comparison: Tanezumab 5 mg vs Celecoxib; Week 24: >=30%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = 12.0, 95% CI 2-sided [-2.3 to 25.7]
Statistical Analysis 10: Comparison: Tanezumab 10 mg vs Celecoxib; Week 24: >=30%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = -1.6, 95% CI 2-sided [-15.9 to 12.6]
Statistical Analysis 11: Comparison: Tanezumab 5 mg vs Celecoxib; Week 24: >=50%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = 12.0, 95% CI 2-sided [-2.4 to 25.8]
Statistical Analysis 12: Comparison: Tanezumab 10 mg vs Celecoxib; Week 24: >=50%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = 5.0, 95% CI 2-sided [-9.1 to 18.9]
Statistical Analysis 13: Comparison: Tanezumab 5 mg vs Celecoxib; Week 24: >=70%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = 14.1, 95% CI 2-sided [2.9 to 24.8]
Statistical Analysis 14: Comparison: Tanezumab 10 mg vs Celecoxib; Week 24: >=70%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = 10.6, 95% CI 2-sided [-0.2 to 21.0]
Statistical Analysis 15: Comparison: Tanezumab 5 mg vs Celecoxib; Week 24: >=90%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = 5.4, 95% CI 2-sided [-0.7 to 11.4]
Statistical Analysis 16: Comparison: Tanezumab 10 mg vs Celecoxib; Week 24: >=90%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = 3.2, 95% CI 2-sided [-2.2 to 8.5]
Statistical Analysis 17: Comparison: Tanezumab 5 mg vs Celecoxib; Week 40: >=30%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = 17.4, 95% CI 2-sided [3.1 to 30.9]
Statistical Analysis 18: Comparison: Tanezumab 10 mg vs Celecoxib; Week 40: >=30%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = -0.5, 95% CI 2-sided [-14.8 to 13.7]
Statistical Analysis 19: Comparison: Tanezumab 5 mg vs Celecoxib; Week 40: >=50%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = 17.4, 95% CI 2-sided [3.0 to 31.0]
Statistical Analysis 20: Comparison: Tanezumab 10 mg vs Celecoxib; Week 40: >=50%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = 5.0, 95% CI 2-sided [-9.0 to 18.7]
Statistical Analysis 21: Comparison: Tanezumab 5 mg vs Celecoxib; Week 40: >=70%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = 17.4, 95% CI 2-sided [4.6 to 29.4]
Statistical Analysis 22: Comparison: Tanezumab 10 mg vs Celecoxib; Week 40: >=70%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = 7.3, 95% CI 2-sided [-4.5 to 18.9]
Statistical Analysis 23: Comparison: Tanezumab 5 mg vs Celecoxib; Week 40: >=90%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = 7.6, 95% CI 2-sided [1.4 to 13.5]
Statistical Analysis 24: Comparison: Tanezumab 10 mg vs Celecoxib; Week 40: >=90%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = 5.4, 95% CI 2-sided [-0.1 to 10.6]
Statistical Analysis 25: Comparison: Tanezumab 5 mg vs Celecoxib; Week 56: >=30%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = 12.0, 95% CI 2-sided [-2.4 to 25.8]
Statistical Analysis 26: Comparison: Tanezumab 10 mg vs Celecoxib; Week 56: >=30%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = -3.8, 95% CI 2-sided [-17.9 to 10.5]
Statistical Analysis 27: Comparison: Tanezumab 5 mg vs Celecoxib; Week 56: >=50%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = 12.0, 95% CI 2-sided [-2.5 to 25.9]
Statistical Analysis 28: Comparison: Tanezumab 10 mg vs Celecoxib; Week 56: >=50%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = -2.6, 95% CI 2-sided [-16.5 to 11.4]
Statistical Analysis 29: Comparison: Tanezumab 5 mg vs Celecoxib; Week 56: >=70%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = 18.5, 95% CI 2-sided [5.6 to 30.5]
Statistical Analysis 30: Comparison: Tanezumab 10 mg vs Celecoxib; Week 56: >=70%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = 8.4, 95% CI 2-sided [-3.6 to 20.0]
Statistical Analysis 31: Comparison: Tanezumab 5 mg vs Celecoxib; Week 56: >=90%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = 8.7, 95% CI 2-sided [1.6 to 15.4]
Statistical Analysis 32: Comparison: Tanezumab 10 mg vs Celecoxib; Week 56: >=90%; Test type: Other — No formal hypotheses were tested in the study; Difference in Percentage of Participants = 3.2, 95% CI 2-sided [-2.2 to 8.5]

36. Secondary Outcome: Change From Baseline in Brief Pain Inventory-short Form (BPI-sf) Scores for Worst Pain at Weeks 2, 4, 8, 16, 24, 40, 56, and 64
Description: BPI-sf is a self-administered questionnaire to assess the severity of pain and pain interference on daily functions during 24 hours prior to evaluation at specified time points. BPI-sf scores for worst pain: participants were asked to rate their pain by circling any 1 number from 0 (no pain) to 10 (pain as bad as you can imagine) that best describes their pain at its worst in the last 24 hours; higher scores indicated worse pain.
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 40, 56 and 64
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
units on a scale
  Change at Week 2 | -0.82 (1.26) | -0.81 (1.67) | -0.61 (1.48)
  Change at Week 4: number analyzed (Participants) | 92 | 92 | 91
  Change at Week 4 | -1.25 (1.82) | -1.22 (1.89) | -0.95 (1.68)
  Change at Week 8: number analyzed (Participants) | 92 | 92 | 90
  Change at Week 8 | -1.65 (1.97) | -1.89 (2.18) | -1.28 (1.69)
  Change at Week 16: number analyzed (Participants) | 91 | 89 | 88
  Change at Week 16 | -3.26 (2.03) | -2.92 (2.32) | -2.67 (2.13)
  Change at Week 24: number analyzed (Participants) | 63 | 50 | 48
  Change at Week 24 | -4.27 (1.99) | -4.78 (1.81) | -4.13 (1.79)
  Change at Week 40: number analyzed (Participants) | 63 | 44 | 44
  Change at Week 40 | -4.70 (1.85) | -4.64 (1.59) | -4.39 (1.85)
  Change at Week 56: number analyzed (Participants) | 63 | 43 | 43
  Change at Week 56 | -4.76 (1.96) | -4.70 (2.03) | -4.47 (1.91)
  Change at Week 64: number analyzed (Participants) | 62 | 43 | 43
  Change at Week 64 | -3.71 (2.25) | -3.51 (1.99) | -3.91 (2.28)

37. Secondary Outcome: Change From Baseline in Brief Pain Inventory-short Form (BPI-sf) Scores for Average Pain at Weeks 2, 4, 8, 16, 24, 40, 56, and 64
Description: BPI-sf is a self-administered questionnaire to assess the severity of pain and pain interference on daily functions during 24 hours prior to evaluation at specified/scheduled time points. BPI-sf scores for average pain: participants were asked to rate their pain by circling any 1 number from 0 (no pain) to 10 (pain as bad as you can imagine) that best describes their pain on average in the last 24 hours; higher scores indicated worse pain.
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 40, 56 and 64
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
units on a scale
  Change at Week 2 | -0.68 (1.35) | -0.78 (1.44) | -0.50 (1.36)
  Change at Week 4: number analyzed (Participants) | 92 | 92 | 91
  Change at Week 4 | -1.12 (1.75) | -1.28 (1.72) | -1.01 (1.43)
  Change at Week 8: number analyzed (Participants) | 92 | 92 | 90
  Change at Week 8 | -1.49 (1.84) | -1.87 (1.99) | -1.16 (1.73)
  Change at Week 16: number analyzed (Participants) | 91 | 89 | 88
  Change at Week 16 | -3.07 (2.03) | -3.07 (2.03) | -2.57 (1.89)
  Change at Week 24: number analyzed (Participants) | 63 | 50 | 48
  Change at Week 24 | -4.10 (1.73) | -4.66 (1.52) | -3.92 (1.66)
  Change at Week 40: number analyzed (Participants) | 63 | 44 | 44
  Change at Week 40 | -4.38 (1.46) | -4.50 (1.39) | -4.16 (1.61)
  Change at Week 56: number analyzed (Participants) | 63 | 43 | 43
  Change at Week 56 | -4.43 (1.70) | -4.42 (1.59) | -4.30 (1.63)
  Change at Week 64: number analyzed (Participants) | 62 | 43 | 43
  Change at Week 64 | -3.53 (1.93) | -3.72 (1.62) | -3.70 (1.91)

38. Secondary Outcome: Change From Baseline in Brief Pain Inventory-short Form (BPI-sf) Scores for Pain Interference Index at Weeks 2, 4, 8, 16, 24, 40, 56, and 64
Description: BPI-sf is a self-administered questionnaire to assess the severity of pain and pain interference on daily functions during 24 hours prior to evaluation at specified/scheduled time points. Pain interference index was calculated as the mean of the 7 BPI-sf pain interference items: pain interference with general activity; mood; walking ability; normal work (outside home and housework); relations with other people; sleep and enjoyment of life. Each of the 7 items had score range from 0 (does not interfere) to 10 (completely interferes), higher scores indicated more interference in daily activities due to pain. Overall score range for pain interference index was 0 (no interference) to 10 (complete interference), higher score = higher interference.
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 40, 56 and 64
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or matching placebo). Here, 'Number Analyzed' = participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
units on a scale
  Change at Week 2 | -0.98 (1.76) | -0.87 (1.51) | -0.78 (1.94)
  Change at Week 4: number analyzed (Participants) | 92 | 92 | 91
  Change at Week 4 | -1.43 (1.94) | -1.32 (1.74) | -1.16 (1.92)
  Change at Week 8: number analyzed (Participants) | 92 | 92 | 90
  Change at Week 8 | -1.75 (1.99) | -1.84 (1.93) | -1.51 (2.14)
  Change at Week 16: number analyzed (Participants) | 91 | 89 | 88
  Change at Week 16 | -2.98 (2.10) | -2.70 (2.13) | -2.62 (2.39)
  Change at Week 24: number analyzed (Participants) | 63 | 50 | 48
  Change at Week 24 | -3.76 (2.07) | -3.74 (2.02) | -3.52 (1.97)
  Change at Week 40: number analyzed (Participants) | 63 | 44 | 44
  Change at Week 40 | -3.88 (1.92) | -3.48 (2.02) | -3.69 (2.03)
  Change at Week 56: number analyzed (Participants) | 63 | 43 | 43
  Change at Week 56 | -3.86 (2.09) | -3.79 (1.95) | -3.54 (2.25)
  Change at Week 64: number analyzed (Participants) | 62 | 43 | 43
  Change at Week 64 | -3.31 (2.26) | -3.29 (2.07) | -3.17 (2.42)

39. Secondary Outcome: Change From Baseline in Brief Pain Inventory-short Form (BPI-sf) Scores for Pain Interference With General Activity at Weeks 2, 4, 8, 16, 24, 40, 56, and 64
Description: BPI-sf is a self-administered questionnaire to assess the severity of pain and pain interference on daily functions during 24 hours prior to evaluation at specified/scheduled time points. BPI-sf scores for pain interference with general activity: participants were asked to circle from any 1 number from 0 (no interference) to 10 (complete interference) that described how, during the past 24 hours, pain has interfered with their general activity; higher scores indicated higher interference.
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 40, 56 and 64
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
units on a scale
  Change at Week 2 | -1.10 (1.95) | -1.05 (1.95) | -0.67 (2.20)
  Change at Week 4: number analyzed (Participants) | 92 | 92 | 91
  Change at Week 4 | -1.68 (2.52) | -1.54 (2.26) | -1.26 (2.20)
  Change at Week 8: number analyzed (Participants) | 92 | 92 | 90
  Change at Week 8 | -2.04 (2.44) | -2.04 (2.61) | -1.77 (2.40)
  Change at Week 16: number analyzed (Participants) | 91 | 89 | 88
  Change at Week 16 | -3.29 (2.49) | -3.04 (2.56) | -2.92 (2.45)
  Change at Week 24: number analyzed (Participants) | 63 | 50 | 48
  Change at Week 24 | -4.30 (2.26) | -4.62 (2.00) | -4.06 (2.04)
  Change at Week 40: number analyzed (Participants) | 63 | 44 | 44
  Change at Week 40 | -4.59 (2.07) | -4.36 (2.11) | -4.23 (1.99)
  Change at Week 56: number analyzed (Participants) | 63 | 43 | 43
  Change at Week 56 | -4.49 (2.21) | -4.65 (1.97) | -4.19 (2.21)
  Change at Week 64: number analyzed (Participants) | 62 | 43 | 43
  Change at Week 64 | -3.89 (2.46) | -3.88 (2.33) | -3.63 (2.23)

40. Secondary Outcome: Change From Baseline in Brief Pain Inventory-short Form (BPI-sf) Scores for Pain Interference With Walking Ability at Weeks 2, 4, 8, 16, 24, 40, 56, and 64
Description: BPI-sf is a self-administered questionnaire to assess the severity of pain and pain interference on daily functions during 24 hours prior to evaluation at specified/scheduled time points. BPI-sf scores for pain interference with walking ability: participants were asked to circle from any 1 number from 0 (does not interfere) to 10 (completely interferes) that described how, during the past 24 hours, pain has interfered with their walking ability; higher scores indicated higher interference.
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 40, 56 and 64
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
units on a scale
  Change at Week 2 | -0.89 (2.33) | -1.06 (2.13) | -0.73 (2.26)
  Change at Week 4: number analyzed (Participants) | 92 | 92 | 91
  Change at Week 4 | -1.37 (2.49) | -1.23 (2.35) | -1.12 (2.40)
  Change at Week 8: number analyzed (Participants) | 92 | 92 | 90
  Change at Week 8 | -1.59 (2.41) | -1.91 (2.41) | -1.37 (2.54)
  Change at Week 16: number analyzed (Participants) | 91 | 89 | 88
  Change at Week 16 | -2.89 (2.53) | -2.60 (2.63) | -2.52 (2.86)
  Change at Week 24: number analyzed (Participants) | 63 | 50 | 48
  Change at Week 24 | -3.81 (2.51) | -3.76 (2.40) | -3.44 (2.01)
  Change at Week 40: number analyzed (Participants) | 63 | 44 | 44
  Change at Week 40 | -3.78 (2.30) | -3.36 (2.26) | -3.64 (2.04)
  Change at Week 56: number analyzed (Participants) | 63 | 43 | 43
  Change at Week 56 | -3.76 (2.39) | -3.58 (2.37) | -3.56 (2.28)
  Change at Week 64: number analyzed (Participants) | 62 | 43 | 43
  Change at Week 64 | -3.18 (2.53) | -3.09 (2.45) | -3.16 (2.53)

41. Secondary Outcome: Change From Baseline in Brief Pain Inventory-short Form (BPI-sf) Scores for Pain Interference With Sleep at Weeks 2, 4, 8, 16, 24, 40, 56, and 64
Description: BPI-sf is a self-administered questionnaire to assess the severity of pain and pain interference on daily functions during 24 hours prior to evaluation at specified/scheduled time points. BPI-sf scores for pain interference with sleep: participants were asked to circle from any 1 number from 0 (does not interfere) to 10 (completely interferes) that described how, during the past 24 hours, pain has interfered with their sleep; higher scores indicated higher interference.
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 40, 56 and 64
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
units on a scale
  Change at Week 2 | -1.02 (2.57) | -0.77 (2.34) | -0.59 (2.37)
  Change at Week 4: number analyzed (Participants) | 92 | 92 | 91
  Change at Week 4 | -1.28 (2.54) | -1.37 (2.32) | -0.85 (2.57)
  Change at Week 8: number analyzed (Participants) | 92 | 92 | 90
  Change at Week 8 | -1.80 (2.64) | -1.96 (2.45) | -1.29 (2.44)
  Change at Week 16: number analyzed (Participants) | 91 | 89 | 88
  Change at Week 16 | -2.97 (2.58) | -2.75 (2.69) | -2.30 (2.89)
  Change at Week 24: number analyzed (Participants) | 63 | 50 | 48
  Change at Week 24 | -3.62 (2.55) | -3.46 (2.73) | -3.19 (2.74)
  Change at Week 40: number analyzed (Participants) | 63 | 44 | 44
  Change at Week 40 | -3.73 (2.48) | -3.25 (2.82) | -3.41 (2.71)
  Change at Week 56: number analyzed (Participants) | 63 | 43 | 43
  Change at Week 56 | -3.78 (2.60) | -3.65 (2.92) | -3.19 (2.91)
  Change at Week 64: number analyzed (Participants) | 62 | 43 | 43
  Change at Week 64 | -3.26 (2.73) | -3.35 (2.80) | -2.79 (3.09)

42. Secondary Outcome: Change From Baseline in Brief Pain Inventory-short Form (BPI-sf) Scores for Pain Interference With Normal Work at Weeks 2, 4, 8, 16, 24, 40, 56 and 64
Description: BPI-sf is a self-administered questionnaire to assess the severity of pain and pain interference on daily functions during 24 hours prior to evaluation at specified/scheduled time points. BPI-sf scores for pain interference with normal work: participants were asked to circle from any 1 number from 0 (does not interfere) to 10 (completely interferes) that described how, during the past 24 hours, pain has interfered with their normal work; higher scores indicated higher interference.
Time Frame: Baseline, Weeks 2, 4, 8, 16, 24, 40, 56 and 64
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
units on a scale
  Change at Week 2 | -1.04 (2.44) | -1.17 (2.28) | -0.96 (2.33)
  Change at Week 4: number analyzed (Participants) | 92 | 92 | 91
  Change at Week 4 | -1.49 (2.39) | -1.39 (2.29) | -1.30 (2.27)
  Change at Week 8: number analyzed (Participants) | 92 | 92 | 90
  Change at Week 8 | -1.93 (2.55) | -2.11 (2.49) | -1.69 (2.43)
  Change at Week 16: number analyzed (Participants) | 91 | 89 | 88
  Change at Week 16 | -3.35 (2.71) | -3.04 (2.68) | -2.93 (2.74)
  Change at Week 24: number analyzed (Participants) | 63 | 50 | 48
  Change at Week 24 | -4.44 (2.58) | -4.26 (2.51) | -4.02 (2.15)
  Change at Week 40: number analyzed (Participants) | 63 | 44 | 44
  Change at Week 40 | -4.52 (2.33) | -3.86 (2.29) | -4.16 (2.52)
  Change at Week 56: number analyzed (Participants) | 63 | 43 | 43
  Change at Week 56 | -4.49 (2.78) | -4.16 (2.35) | -4.14 (2.36)
  Change at Week 64: number analyzed (Participants) | 62 | 43 | 43
  Change at Week 64 | -3.84 (2.81) | -3.53 (2.59) | -3.77 (2.58)

43. Secondary Outcome: Percentage of Participants With Chronic Low Back Pain Responders Index at Weeks 16, 24, 40 and 56
Description: Chronic low back pain responder index analysis is a composite endpoint of average low back pain intensity (aLBPI) score, PGA of low back pain, and RMDQ total score. aLBPI: evaluate average pain during the past 24 hours, range 0 (no pain) to 10 (worst possible pain), higher scores = higher worse pain. PGA of low back pain: evaluated participants' well-being due to low back pain on day of assessment, range 1 (very good) to 5 (very poor), higher scores = worse condition. RMDQ total score: assessed ability to perform daily activities, range 0 (no disability) to 24 (maximum disability), higher scores = more disability. Participants were successful responders if they had: >=30 percent reduction in aLBPI from baseline to particular week; decrease of >=30 percent in PGA of low back pain from baseline to particular week and no worsening (increase) in RMDQ total score from baseline to particular week.
Time Frame: Weeks 16, 24, 40 and 56
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or placebo matched to tanezumab). Number Analyzed = participants evaluable for this outcome measure at specified time points.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
percentage of participants
  Week 16 | 54.3 [44.2 to 64.1] | 48.4 [38.5 to 58.4] | 50.0 [40.0 to 60.0]
  Week 24 | 53.3 [43.1 to 63.1] | 45.2 [35.4 to 55.3] | 42.4 [32.8 to 52.6]
  Week 40 | 56.5 [46.3 to 66.2] | 43.0 [33.4 to 53.2] | 41.3 [31.8 to 51.5]
  Week 56 | 51.1 [41.0 to 61.1] | 39.8 [30.4 to 50.0] | 42.4 [32.8 to 52.6]

44. Secondary Outcome: Percentage of Participants Achieving Change of >=2 Points From Baseline in Patient's Global Assessment (PGA) of Low Back Pain at Weeks 16, 24, 40 and 56
Description: PGA of low back pain assessed by asking question to participants: "Considering all ways your low back pain affects you, how are you doing today?" They responded on 5 point Likert scale ranging from 1 to 5, using IRT, where 1= very good (asymptomatic and no limitation of normal activities); 2= good (mild symptoms and no limitation of normal activities); 3= fair (moderate symptoms and limitation of some normal activities); 4= poor (severe symptoms and inability to carry out most normal activities); 5= very poor (very severe symptoms which are intolerable and inability to carry out all normal activities). Higher scores indicated worsening of condition. Percentage of participants with positive change of at least 2 points from baseline in PGA of low back pain were reported.
Time Frame: Baseline, Weeks 16, 24, 40 and 56
Population: as for outcome 34
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
percentage of participants
  Week 16 | 17.4 [10.9 to 26.5] | 12.9 [7.4 to 21.4] | 16.3 [10.0 to 25.3]
  Week 24 | 18.5 [11.8 to 27.7] | 15.1 [9.1 to 23.8] | 9.8 [5.0 to 17.8]
  Week 40 | 23.9 [16.3 to 33.6] | 11.8 [6.6 to 20.1] | 9.8 [5.0 to 17.8]
  Week 56 | 18.5 [11.8 to 27.7] | 11.8 [6.6 to 20.1] | 10.9 [5.8 to 19.0]

45. Secondary Outcome: European Quality of Life-5 Dimension-5 Levels (EQ-5D-5L): Dimensions Scores at Baseline, Weeks 16 and 56
Description: EQ-5D-5L is a standardized participant completed questionnaire that measures health-related quality of life and translates that score into an index value or utility score. EQ-5D-5L consists of two components: a health state profile and an optional visual analogue scale (VAS). EQ-5D health state profile is comprised of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1= no problems, 2= slight problems, 3= moderate problems, 4= severe problems, and 5= extreme problems. Higher scores indicated greater levels of problems across each of the five dimensions.
Time Frame: Baseline, Weeks 16 and 56
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or placebo matched to tanezumab). Here, 'Number Analyzed' = Participants evaluable for this outcome measure for specified rows.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
units on a scale
  Baseline: Mobility | 2.3 (0.78) | 2.2 (0.95) | 2.3 (0.97)
  Baseline: Self-care | 1.8 (0.81) | 1.6 (0.82) | 1.6 (0.81)
  Baseline: Usual activities | 2.4 (0.83) | 2.4 (0.83) | 2.3 (0.79)
  Baseline: Pain/Discomfort | 2.9 (0.69) | 2.9 (0.71) | 2.9 (0.64)
  Baseline: Anxiety/Depression | 1.8 (0.83) | 1.8 (0.97) | 1.6 (0.81)
  Week 16: Mobility: number analyzed (Participants) | 92 | 90 | 88
  Week 16: Mobility | 1.6 (0.77) | 1.5 (0.80) | 1.5 (0.77)
  Week 16: Self-care: number analyzed (Participants) | 92 | 90 | 88
  Week 16: Self-care | 1.2 (0.48) | 1.1 (0.35) | 1.2 (0.48)
  Week 16: Usual activities: number analyzed (Participants) | 92 | 90 | 88
  Week 16: Usual activities | 1.6 (0.71) | 1.5 (0.66) | 1.6 (0.69)
  Week 16: Pain/Discomfort: number analyzed (Participants) | 92 | 90 | 88
  Week 16: Pain/Discomfort | 2.0 (0.74) | 2.0 (0.75) | 2.1 (0.67)
  Week 16: Anxiety/Depression: number analyzed (Participants) | 92 | 90 | 88
  Week 16: Anxiety/Depression | 1.2 (0.59) | 1.2 (0.52) | 1.2 (0.47)
  Week 56: Mobility: number analyzed (Participants) | 63 | 43 | 43
  Week 56: Mobility | 1.3 (0.55) | 1.3 (0.54) | 1.4 (0.73)
  Week 56: Self-care: number analyzed (Participants) | 63 | 43 | 43
  Week 56: Self-care | 1.0 (0.21) | 1.1 (0.26) | 1.0 (0.15)
  Week 56: Usual activities: number analyzed (Participants) | 63 | 43 | 43
  Week 56: Usual activities | 1.3 (0.46) | 1.3 (0.50) | 1.3 (0.51)
  Week 56: Pain/Discomfort: number analyzed (Participants) | 63 | 43 | 43
  Week 56: Pain/Discomfort | 1.7 (0.63) | 1.7 (0.59) | 1.8 (0.55)
  Week 56: Anxiety/Depression: number analyzed (Participants) | 63 | 43 | 43
  Week 56: Anxiety/Depression | 1.1 (0.56) | 1.1 (0.29) | 1.1 (0.26)

46. Secondary Outcome: European Quality of Life-5 Dimension-5 Levels (EQ-5D-5L): Overall Health Utility Score/ Index Value
Description: EQ-5D health state profile has 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: 1= no problems, 2= slight problems, 3= moderate problems, 4= severe problems, and 5= extreme problems. Responses from each of the 5 domains were used to calculate overall health state/a single utility index value. Example: if a participant responded "no problems" for each 5 dimensions, then health state was coded as "11111" with a predefined single index value to it. Every health state (coded as combination of responses on each of 5 dimensions) had a unique predefined utility index value assigned to it, by EuroQol. Japan value sets (with all possible health states) was used in the study, overall health utility score ranged from -0.111 (minimum score) to 1 (maximum score). Higher (positive) scores = better health state.
Time Frame: Baseline, Weeks 16 and 56
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
units on a scale
  Baseline | 0.61 (0.09) | 0.62 (0.11) | 0.63 (0.09)
  Week 16: number analyzed (Participants) | 92 | 90 | 88
  Week 16 | 0.76 (0.14) | 0.77 (0.13) | 0.76 (0.13)
  Week 56: number analyzed (Participants) | 63 | 43 | 43
  Week 56 | 0.83 (0.13) | 0.83 (0.13) | 0.82 (0.12)

47. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment Questionnaire: Low Back Pain (WPAI:LBP)- Percent Work Time Missed Due to Chronic Low Back Pain at Weeks 16, 56 and 64
Description: WPAI:LBP is a participant rated questionnaire that measures the effect of participant's chronic low back pain (CLBP) on general health and symptom severity on work productivity and regular activities. Percentage of work time missed by participants due to CLBP was recorded on a score range of 0 (no impact on work time) to 100 (extreme impact on work time), higher scores indicated greater work time missed and lesser productivity.
Time Frame: Baseline, Weeks 16, 56 and 64
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: percentage of work time missed
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
percentage of work time missed
  Baseline: number analyzed (Participants) | 71 | 68 | 58
  Baseline | 5.0 (17.40) | 5.7 (16.91) | 5.8 (18.74)
  Change at Week 16: number analyzed (Participants) | 64 | 65 | 53
  Change at Week 16 | -0.8 (12.53) | -4.8 (15.11) | -1.9 (14.04)
  Change at Week 56: number analyzed (Participants) | 47 | 32 | 28
  Change at Week 56 | -2.4 (7.15) | -2.3 (10.47) | -1.3 (4.13)
  Change at Week 64: number analyzed (Participants) | 42 | 31 | 26
  Change at Week 64 | -1.6 (6.67) | -0.6 (6.37) | 3.1 (16.20)

48. Secondary Outcome: Change From Baseline in in Work Productivity and Activity Impairment Questionnaire: Low Back Pain (WPAI:LBP)- Percent Impairment While Working Due to Chronic Low Back Pain at Weeks 16, 56 and 64
Description: WPAI: LBP is a participant rated questionnaire that measures the effect of participant's chronic low back pain (CLBP) on general health and symptom severity on work productivity and regular activities. Percentage of impairment while working due to CLBP was recorded on a score range of 0 (no impairment) to 100 (extreme impairment), higher scores indicated greater impairment while working and lesser productivity.
Time Frame: Baseline, Weeks 16, 56 and 64
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: percentage of impairment
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
percentage of impairment
  Baseline: number analyzed (Participants) | 69 | 67 | 56
  Baseline | 55.4 (24.29) | 53.7 (24.97) | 56.4 (22.03)
  Change at Week 16: number analyzed (Participants) | 64 | 64 | 52
  Change at Week 16 | -31.6 (26.68) | -24.7 (30.29) | -28.3 (25.57)
  Change at Week 56: number analyzed (Participants) | 47 | 32 | 28
  Change at Week 56 | -38.7 (24.99) | -36.6 (28.69) | -27.1 (26.23)
  Change at Week 64: number analyzed (Participants) | 42 | 31 | 26
  Change at Week 64 | -31.9 (23.19) | -33.9 (28.01) | -30.8 (25.91)

49. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment Questionnaire: Low Back Pain (WPAI:LBP)- Percent Overall Work Impairment Due to Chronic Low Back Pain at Weeks 16, 56 and 64
Description: WPAI: LBP is a participant rated questionnaire that measures the effect of participant's chronic low back pain (CLBP) on general health and symptom severity on work productivity and regular activities. Percentage of overall work impairment due to CLBP was recorded on a score range of 0 (no impairment) to 100 (extreme impairment), higher scores indicated greater overall work impairment and lesser productivity.
Time Frame: Baseline, Weeks 16, 56 and 64
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: percentage of impairment
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
percentage of impairment
  Baseline: number analyzed (Participants) | 69 | 67 | 56
  Baseline | 56.0 (24.65) | 56.0 (24.38) | 57.2 (22.26)
  Change at Week 16: number analyzed (Participants) | 64 | 64 | 52
  Change at Week 16 | -31.8 (27.33) | -26.8 (29.90) | -27.8 (27.29)
  Change at Week 56: number analyzed (Participants) | 47 | 32 | 28
  Change at Week 56 | -39.2 (25.51) | -38.3 (28.98) | -27.7 (25.76)
  Change at Week 64: number analyzed (Participants) | 42 | 31 | 26
  Change at Week 64 | -32.1 (23.44) | -33.7 (29.52) | -27.9 (26.67)

50. Secondary Outcome: Change From Baseline in Work Productivity and Activity Impairment Questionnaire: Low Back Pain (WPAI:LBP)- Percent Activity Impairment Due to Chronic Low Back Pain at Weeks 16, 56 and 64
Description: WPAI: LBP is a participant rated questionnaire that measures the effect of participant's chronic low back pain (CLBP) on general health and symptom severity on work productivity and regular activities. Percentage of daily activity impairment due to CLBP was recorded on a score range of 0 (no impairment) to 100 (extreme impairment), higher scores indicated greater daily activity impairment and lesser productivity.
Time Frame: Baseline, Weeks 16, 56 and 64
Population: as for outcome 33
Measure: Mean (Standard Deviation); unit: percentage of impairment
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
percentage of impairment
  Baseline | 57.8 (20.10) | 53.7 (22.69) | 54.7 (21.35)
  Change at Week 16: number analyzed (Participants) | 92 | 92 | 91
  Change at Week 16 | -30.1 (24.87) | -25.0 (26.04) | -25.4 (26.13)
  Change at Week 56: number analyzed (Participants) | 63 | 45 | 47
  Change at Week 56 | -42.1 (24.11) | -35.1 (25.19) | -32.6 (23.63)
  Change at Week 64: number analyzed (Participants) | 62 | 43 | 43
  Change at Week 64 | -37.3 (23.27) | -34.4 (23.13) | -33.0 (27.21)

51. Secondary Outcome: Number of Participants Who Discontinued Due to Lack of Efficacy
Description: Number of participants who discontinued from study treatment due to lack of efficacy have been reported here.
Time Frame: Baseline up to Week 56
Population: as for outcome 34
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
Participants | 1 | 4 | 1
Statistical Analysis 1: Comparison: Tanezumab 5 mg vs Celecoxib; 95% CI of proportion is the Agresti-Coull confidence limit; Test type: Other — No formal hypotheses were tested in the study; Difference in proportion = 0, 95% CI 2-sided [-4.1 to 4.1]
Statistical Analysis 2: Comparison: Tanezumab 10 mg vs Celecoxib; 95% CI of proportion is the Agresti-Coull confidence limit; Test type: Other — No formal hypotheses were tested in the study; Difference in proportion = 3.2, 95% CI 2-sided [-2.2 to 8.5]

52. Secondary Outcome: Time to Discontinuation Due to Lack of Efficacy
Description: Time to discontinuation (in days) due to lack of efficacy was defined as the time interval from the date of first study drug administration up to the date of discontinuation of participant from treatment due to lack of efficacy. Results reported below are contributed only by participants who discontinued due to lack of efficacy.
Time Frame: Baseline up to Week 56
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or placebo matched to tanezumab). Participants who discontinued due to lack of efficacy analyzed.
Measure: Number; unit: days
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 1 | 4 | 1
days
  Minimum | 111 | 15 | 141
  1st Percentile | 111 | 15 | 141
  2nd Percentile | NA — Cannot be estimated using Kaplan-Meier method due to an insufficient number of participants with events. | 29 | 141
  5th Percentile | NA — Cannot be estimated using Kaplan-Meier method due to an insufficient number of participants with events. | NA — Cannot be estimated using Kaplan-Meier method due to an insufficient number of participants with events. | NA — Cannot be estimated using Kaplan-Meier method due to an insufficient number of participants with events.
  Maximum | 111 | 113 | 141

53. Secondary Outcome: Number of Participants Who Took Rescue Medication During Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48, 56 and 64: Observed Data
Description: In case of inadequate pain relief, acetaminophen/paracetamol tablets up to 3000 mg per day up to 3 days in a week could be taken as rescue medication between Day 1 to Week 64. Number of participants with any use of rescue medication during each specified/scheduled study week were summarized.
Time Frame: Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48, 56 and 64
Population: ITT population was analyzed. Here, 'Number Analyzed' = participants evaluable for this outcome measure at specified time points. Observed data: analysis was performed using all available data at specified weeks and no imputation technique was used for missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
Participants
  Week 2 | 36 | 24 | 33
  Week 4: number analyzed (Participants) | 92 | 93 | 91
  Week 4 | 30 | 23 | 27
  Week 8: number analyzed (Participants) | 92 | 91 | 90
  Week 8 | 28 | 19 | 25
  Week 12: number analyzed (Participants) | 91 | 89 | 90
  Week 12 | 17 | 14 | 27
  Week 16: number analyzed (Participants) | 91 | 88 | 88
  Week 16 | 14 | 18 | 21
  Week 24: number analyzed (Participants) | 68 | 57 | 54
  Week 24 | 21 | 10 | 14
  Week 32: number analyzed (Participants) | 63 | 48 | 46
  Week 32 | 14 | 9 | 12
  Week 40: number analyzed (Participants) | 63 | 45 | 45
  Week 40 | 11 | 10 | 5
  Week 48: number analyzed (Participants) | 63 | 45 | 44
  Week 48 | 15 | 9 | 8
  Week 56: number analyzed (Participants) | 63 | 43 | 43
  Week 56 | 16 | 9 | 9
  Week 64: number analyzed (Participants) | 61 | 45 | 44
  Week 64 | 23 | 13 | 14

54. Secondary Outcome: Number of Participants Who Took Rescue Medication During Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48 and 56: Last Observation Carried Forward (LOCF)
Description: In case of inadequate pain relief, acetaminophen/paracetamol caplets, tablets, or capsules up to 3000 mg per day up to 3 days in a week could be taken as rescue medication between Day 1 to Week 64. Number of participants with any use of rescue medication during each specified/scheduled study week were summarized.
Time Frame: Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48 and 56
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or placebo matched to tanezumab). Last observation was carried forward for missing data.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
Participants
  Week 2 | 37 | 24 | 33
  Week 4 | 30 | 24 | 28
  Week 8 | 28 | 19 | 27
  Week 12 | 17 | 16 | 29
  Week 16 | 15 | 21 | 26
  Week 24 | 32 | 26 | 32
  Week 32 | 27 | 27 | 34
  Week 40 | 24 | 30 | 27
  Week 48 | 28 | 28 | 30
  Week 56 | 29 | 28 | 32

55. Secondary Outcome: Number of Days of Rescue Medication Use During Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48, 56 and 64: Observed Data
Description: In case of inadequate pain relief, acetaminophen/paracetamol tablets up to 3000 mg per day up to 3 days in a week could be taken as rescue medication between Day 1 to Week 64. Number of days the participants used the rescue medication during each specified/scheduled study week were summarized.
Time Frame: Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48, 56 and 64
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
days
  Week 2 | 0.9 (1.37) | 0.8 (1.57) | 0.8 (1.35)
  Week 4: number analyzed (Participants) | 92 | 93 | 91
  Week 4 | 0.8 (1.29) | 0.6 (1.27) | 0.7 (1.37)
  Week 8: number analyzed (Participants) | 92 | 91 | 90
  Week 8 | 0.6 (1.08) | 0.4 (0.92) | 0.7 (1.22)
  Week 12: number analyzed (Participants) | 91 | 89 | 90
  Week 12 | 0.4 (0.98) | 0.4 (1.14) | 0.7 (1.34)
  Week 16: number analyzed (Participants) | 91 | 88 | 88
  Week 16 | 0.5 (1.15) | 0.4 (0.95) | 0.5 (1.10)
  Week 24: number analyzed (Participants) | 68 | 57 | 54
  Week 24 | 1.1 (2.14) | 0.4 (1.41) | 1.0 (2.10)
  Week 32: number analyzed (Participants) | 63 | 48 | 46
  Week 32 | 0.7 (1.75) | 0.3 (1.14) | 0.7 (1.79)
  Week 40: number analyzed (Participants) | 63 | 45 | 45
  Week 40 | 0.5 (1.46) | 0.5 (1.27) | 0.5 (1.63)
  Week 48: number analyzed (Participants) | 63 | 45 | 44
  Week 48 | 0.8 (1.84) | 0.4 (1.17) | 0.6 (1.72)
  Week 56: number analyzed (Participants) | 63 | 43 | 43
  Week 56 | 0.7 (1.69) | 0.4 (1.26) | 0.4 (1.50)
  Week 64: number analyzed (Participants) | 61 | 45 | 44
  Week 64 | 1.1 (1.89) | 0.6 (1.54) | 1.0 (2.08)

56. Secondary Outcome: Number of Days of Rescue Medication Use During Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48 and 56: LOCF
Description: In case of inadequate pain relief, acetaminophen/paracetamol caplets, tablets, or capsules up to 3000 mg per day up to 3 days in a week could be taken as rescue medication between Day 1 to Week 64. Number of days the participants used the rescue medication during each specified/scheduled study week were summarized.
Time Frame: Weeks 2, 4, 8, 12, 16, 24, 32, 40, 48 and 56
Population: as for outcome 54
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
days
  Week 2 | 1.0 (1.37) | 0.8 (1.57) | 0.8 (1.35)
  Week 4 | 0.8 (1.29) | 0.6 (1.27) | 0.8 (1.40)
  Week 8 | 0.6 (1.08) | 0.4 (0.95) | 0.8 (1.43)
  Week 12 | 0.4 (0.98) | 0.5 (1.18) | 0.8 (1.56)
  Week 16 | 0.5 (1.24) | 0.6 (1.47) | 0.7 (1.46)
  Week 24 | 1.5 (2.49) | 1.2 (2.36) | 1.6 (2.66)
  Week 32 | 1.3 (2.43) | 1.2 (2.36) | 1.5 (2.58)
  Week 40 | 1.2 (2.34) | 1.3 (2.35) | 1.4 (2.56)
  Week 48 | 1.3 (2.46) | 1.2 (2.35) | 1.5 (2.56)
  Week 56 | 1.3 (2.41) | 1.3 (2.36) | 1.4 (2.52)

57. Secondary Outcome: Amount of Rescue Medication Used in Weeks 2, 4, 8, 12, and 16: Observed Data
Description: In case of inadequate pain relief, acetaminophen/paracetamol tablets up to 3000 mg per day up to 3 days in a week could be taken as rescue medication between Day 1 to Week 64. Amount of rescue medication used during each specified/scheduled study week were summarized.
Time Frame: Weeks 2, 4, 8, 12 and 16
Population: as for outcome 53
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
milligrams
  Week 2 | 1029 (2118) | 701 (1710) | 809 (1789)
  Week 4: number analyzed (Participants) | 92 | 92 | 91
  Week 4 | 885 (1913) | 440 (1125) | 812 (1744)
  Week 8: number analyzed (Participants) | 92 | 90 | 89
  Week 8 | 813 (1792) | 559 (1577) | 776 (1805)
  Week 12: number analyzed (Participants) | 91 | 87 | 89
  Week 12 | 655 (1845) | 477 (1674) | 657 (1585)
  Week 16: number analyzed (Participants) | 80 | 79 | 77
  Week 16 | 680 (1850) | 292 (1135) | 642 (1810)

58. Secondary Outcome: Amount of Rescue Medication Used in Weeks 2, 4, 8, 12, and 16: LOCF
Description: In case of inadequate pain relief, acetaminophen/paracetamol caplets, tablets, or capsules up to 3000 mg per day up to 3 days in a week could be taken as rescue medication between Day 1 to Week 64. Amount of rescue medication used during each specified/scheduled study week were summarized.
Time Frame: Weeks 2, 4, 8, 12 and 16
Population: as for outcome 54
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
milligrams
  Week 2 | 1042 (2115) | 701 (1710) | 809 (1789)
  Week 4 | 885 (1913) | 543 (1428) | 821 (1737)
  Week 8 | 813 (1792) | 661 (1806) | 855 (1900)
  Week 12 | 648 (1837) | 631 (1956) | 742 (1710)
  Week 16 | 693 (1847) | 584 (1919) | 652 (1800)

59. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Visits of Services Received Directly Related to Low Back Pain
Description: Low back pain HCRU assessed utilization of healthcare resources usage during last 3 months (last 3 months before Baseline [Day 1] visit, weeks 64 and 80 visit, via IRT). Visits of services directly related to low back pain evaluated were: visits to primary care physician, neurologist, physician assistant or nurse practitioner, pain specialist, orthopedist, physical therapist, chiropractor, alternative medicine or therapy, nutritionist/dietician, radiologist and other practitioner. Participants might have been counted more than once under various rows. Only those rows have been reported which had at least 1 participant evaluable for any reporting arm.
Time Frame: Baseline, Weeks 64 and 80
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or placebo matched to tanezumab). Here, 'Number Analyzed' signifies the number of participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
visits
  Baseline: Primary Care Physician: number analyzed (Participants) | 43 | 37 | 45
  Baseline: Primary Care Physician | 4.9 (11.79) | 3.1 (1.18) | 4.1 (4.77)
  Baseline: Neurologist: number analyzed (Participants) | 1 | 0 | 0
  Baseline: Neurologist | 2.0 |  |
  Baseline:Physician Assistant or Nurse Practitioner: number analyzed (Participants) | 1 | 0 | 0
  Baseline:Physician Assistant or Nurse Practitioner | 3.0 |  |
  Baseline: Pain Specialist: number analyzed (Participants) | 4 | 4 | 4
  Baseline: Pain Specialist | 4.5 (1.00) | 2.8 (0.50) | 5.5 (3.70)
  Baseline: Orthopedist: number analyzed (Participants) | 81 | 79 | 74
  Baseline: Orthopedist | 3.9 (4.83) | 3.3 (1.25) | 3.9 (3.81)
  Baseline: Physical Therapist: number analyzed (Participants) | 11 | 2 | 4
  Baseline: Physical Therapist | 17.5 (22.94) | 3.5 (0.71) | 11.8 (1.26)
  Baseline: Chiropractor: number analyzed (Participants) | 1 | 1 | 2
  Baseline: Chiropractor | 2.0 | 2.0 | 4.0 (4.24)
  Baseline: Alternative Medicine Or Therapy: number analyzed (Participants) | 0 | 2 | 2
  Baseline: Alternative Medicine Or Therapy |  | 13.5 (14.85) | 4.0 (2.83)
  Baseline: Nutritionist/Dietician: number analyzed (Participants) | 0 | 0 | 1
  Baseline: Nutritionist/Dietician |  |  | 1.0
  Baseline: Radiologist: number analyzed (Participants) | 1 | 0 | 0
  Baseline: Radiologist | 1.0 |  |
  Baseline: Other Practitioner: number analyzed (Participants) | 3 | 5 | 8
  Baseline: Other Practitioner | 2.0 (1.00) | 2.6 (1.52) | 8.8 (11.78)
  Week 64: Primary Care Physician: number analyzed (Participants) | 24 | 27 | 25
  Week 64: Primary Care Physician | 4.9 (14.98) | 1.5 (1.25) | 1.8 (1.82)
  Week 64: Neurologist: number analyzed (Participants) | 1 | 0 | 1
  Week 64: Neurologist | 5.0 |  | 1.0
  Week 64: Physician Assistant or Nurse Practitioner: number analyzed (Participants) | 1 | 0 | 0
  Week 64: Physician Assistant or Nurse Practitioner | 2.0 |  |
  Week 64: Pain Specialist: number analyzed (Participants) | 0 | 3 | 4
  Week 64: Pain Specialist |  | 1.7 (0.58) | 2.3 (1.89)
  Week 64: Orthopedist: number analyzed (Participants) | 46 | 48 | 48
  Week 64: Orthopedist | 4.0 (11.33) | 1.8 (1.46) | 4.1 (14.18)
  Week 64: Physical Therapist: number analyzed (Participants) | 4 | 0 | 6
  Week 64: Physical Therapist | 6.5 (3.42) |  | 7.7 (11.31)
  Week 64: Chiropractor: number analyzed (Participants) | 0 | 1 | 0
  Week 64: Chiropractor |  | 6.0 |
  Week 64: Alternative Medicine Or Therapy: number analyzed (Participants) | 1 | 2 | 1
  Week 64: Alternative Medicine Or Therapy | 5.0 | 16.5 (19.09) | 2.0
  Week 64: Podiatrist: number analyzed (Participants) | 0 | 0 | 1
  Week 64: Podiatrist |  |  | 1.0
  Week 64: Radiologist: number analyzed (Participants) | 2 | 0 | 1
  Week 64: Radiologist | 3.0 (2.83) |  | 1.0
  Week 64: Other Practitioner: number analyzed (Participants) | 5 | 5 | 7
  Week 64: Other Practitioner | 3.0 (2.92) | 3.4 (2.51) | 16.3 (36.56)
  Week 80: Primary Care Physician: number analyzed (Participants) | 10 | 5 | 7
  Week 80: Primary Care Physician | 1.5 (0.85) | 1.4 (0.89) | 2.9 (4.49)
  Week 80: Physician Assistant or Nurse Practitioner: number analyzed (Participants) | 1 | 0 | 0
  Week 80: Physician Assistant or Nurse Practitioner | 1.0 |  |
  Week 80: Pain Specialist: number analyzed (Participants) | 1 | 1 | 2
  Week 80: Pain Specialist | 1.0 | 1.0 | 2.0 (0.00)
  Week 80: Orthopedist: number analyzed (Participants) | 26 | 18 | 19
  Week 80: Orthopedist | 2.8 (6.61) | 1.7 (1.28) | 2.6 (3.55)
  Week 80: Physical Therapist: number analyzed (Participants) | 1 | 0 | 1
  Week 80: Physical Therapist | 12.0 |  | 4.0
  Week 80: Chiropractor: number analyzed (Participants) | 0 | 0 | 1
  Week 80: Chiropractor |  |  | 3.0
  Week 80: Alternative Medicine Or Therapy: number analyzed (Participants) | 0 | 0 | 1
  Week 80: Alternative Medicine Or Therapy |  |  | 9.0
  Week 80: Radiologist: number analyzed (Participants) | 1 | 1 | 0
  Week 80: Radiologist | 1.0 | 1.0 |
  Week 80: Other Practitioner: number analyzed (Participants) | 3 | 1 | 3
  Week 80: Other Practitioner | 4.0 (3.61) | 4.0 | 2.3 (1.15)

60. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Participants Visited to the Emergency Room Due to Low Back Pain
Description: Low back pain HCRU assessed utilization of healthcare resources during the last 3 months (last 3 months before Baseline [Day 1] visit, weeks 64 and 80 visit, via IRT). Number of participants who visited the emergency room due to low back pain were evaluated.
Time Frame: Baseline, Weeks 64 and 80
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or placebo matched to tanezumab). Here, 'Number Analyzed' signifies the number of participants who were evaluable at specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
Participants
  Baseline | 0 | 0 | 0
  Week 64: number analyzed (Participants) | 91 | 88 | 84
  Week 64 | 0 | 0 | 2
  Week 80: number analyzed (Participants) | 62 | 42 | 43
  Week 80 | 0 | 0 | 0

61. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Participants Hospitalized Due to Low Back Pain
Description: Low back pain HCRU assessed utilization of healthcare resources during the last 3 months for baseline, weeks 64 and 80, via IRT. Domain evaluated was number of participants who were hospitalized due to low back pain.
Time Frame: Baseline, Weeks 64 and 80
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or placebo matched to tanezumab). Here, "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure. 'Number Analyzed'= Participants who were evaluable at specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 92 | 91
Participants
  Baseline | 0 | 1 | 1
  Week 64: number analyzed (Participants) | 90 | 87 | 85
  Week 64 | 1 | 1 | 1
  Week 80: number analyzed (Participants) | 62 | 42 | 43
  Week 80 | 0 | 0 | 0

62. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Nights Stayed in the Hospital Due to Low Back Pain
Description: Low back pain HCRU assessed utilization of healthcare resources during the last 3 months (last 3 months before Baseline [Day 1] visit, weeks 64 and 80 visit, via IRT). Number of nights stayed in the hospital due to low back pain were evaluated.
Time Frame: Baseline, Weeks 64 and 80
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or placebo matched to tanezumab).Not all participants of the ITT population had data collected at each of time points. Hence, Overall number of participants analyzed=participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: nights
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 1 | 2 | 2
nights
  Baseline: number analyzed (Participants) | 0 | 1 | 1
  Baseline |  | 24.0 [24.0 to 24.0] | 2.0 [2.0 to 2.0]
  Week 64: number analyzed (Participants) | 1 | 1 | 1
  Week 64 | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0] | 2.0 [2.0 to 2.0]
  Week 80: number analyzed (Participants) | 0 | 0 | 0

63. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Participants Who Used Any Aids/Devices for Doing Things
Description: Low back pain HCRU assessed utilization of healthcare resources during the last 3 months (last 3 months before Baseline [Day 1] visit, weeks 64 and 80 visit, via IRT). Number of participants who used any aids/devices for doing things were evaluated. Aids included walking aid, wheelchair, device or utensil for dress/bathe/eat and any other aids/devices.
Time Frame: Baseline, Weeks 64 and 80
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or placebo matched to tanezumab). Here, 'Number Analyzed' = Participants who were evaluable for usage of any aids/devices for doing things at specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
Participants
  Baseline: Walking aid use: Never | 91 | 91 | 90
  Baseline: Walking aid use: Rarely | 1 | 0 | 0
  Baseline: Walking aid use: Sometimes | 0 | 0 | 0
  Baseline: Walking aid use: Often | 0 | 1 | 2
  Baseline: Walking aid use: Always | 0 | 1 | 0
  Baseline: Wheelchair use: Never | 92 | 93 | 92
  Baseline: Wheelchair use: Rarely | 0 | 0 | 0
  Baseline: Wheelchair use: Sometimes | 0 | 0 | 0
  Baseline: Wheelchair use: Often | 0 | 0 | 0
  Baseline: Wheelchair use: Always | 0 | 0 | 0
  Baseline: Device/Utensil to Dress Bathe Eat: Never | 92 | 93 | 91
  Baseline: Device/Utensil to Dress Bathe Eat: Rarely | 0 | 0 | 1
  Baseline: Device/Utensil to Dress Bathe Eat: Sometimes | 0 | 0 | 0
  Baseline: Device/Utensil to Dress Bathe Eat: Often | 0 | 0 | 0
  Baseline: Device/Utensil to Dress Bathe Eat: Always | 0 | 0 | 0
  Baseline: Other Aids or Devices: Never | 90 | 87 | 86
  Baseline: Other Aids or Devices: Rarely | 1 | 1 | 1
  Baseline: Other Aids or Devices: Sometimes | 1 | 2 | 3
  Baseline: Other Aids or Devices: Often | 0 | 2 | 1
  Baseline: Other Aids or Devices: Always | 0 | 1 | 1
  Week 64: Walking aid use: number analyzed (Participants) | 91 | 88 | 86
  Week 64: Walking aid use: Never | 88 | 86 | 85
  Week 64: Walking aid use: Rarely | 1 | 0 | 1
  Week 64: Walking aid use: Sometimes | 2 | 0 | 0
  Week 64: Walking aid use: Often | 0 | 1 | 0
  Week 64: Walking aid use: Always | 0 | 1 | 0
  Week 64: Wheelchair use: number analyzed (Participants) | 91 | 88 | 86
  Week 64: Wheelchair use: Never | 91 | 88 | 86
  Week 64: Wheelchair use: Rarely | 0 | 0 | 0
  Week 64: Wheelchair use: Sometimes | 0 | 0 | 0
  Week 64: Wheelchair use: Often | 0 | 0 | 0
  Week 64: Wheelchair use: Always | 0 | 0 | 0
  Week 64: Device/Utensil to Dress Bathe Eat: number analyzed (Participants) | 91 | 88 | 86
  Week 64: Device/Utensil to Dress Bathe Eat: Never | 91 | 87 | 86
  Week 64: Device/Utensil to Dress Bathe Eat: Rarely | 0 | 0 | 0
  Week 64: Device/Utensil to Dress Bathe Eat: Sometimes | 0 | 0 | 0
  Week 64: Device/Utensil to Dress Bathe Eat: Often | 0 | 1 | 0
  Week 64: Device/Utensil to Dress Bathe Eat: Always | 0 | 0 | 0
  Week 64: Other aids or devices: number analyzed (Participants) | 91 | 88 | 86
  Week 64: Other aids or devices: Never | 88 | 85 | 80
  Week 64: Other aids or devices: Rarely | 0 | 1 | 2
  Week 64: Other aids or devices: Sometimes | 1 | 2 | 1
  Week 64: Other aids or devices: Often | 2 | 0 | 1
  Week 64: Other aids or devices: Always | 0 | 0 | 2
  Week 80: Walking aid use: number analyzed (Participants) | 62 | 42 | 43
  Week 80: Walking aid use: Never | 61 | 41 | 42
  Week 80: Walking aid use: Rarely | 1 | 1 | 0
  Week 80: Walking aid use: Sometimes | 0 | 0 | 1
  Week 80: Walking aid use: Often | 0 | 0 | 0
  Week 80: Walking aid use: Always | 0 | 0 | 0
  Week 80: Wheelchair use: number analyzed (Participants) | 62 | 42 | 43
  Week 80: Wheelchair use: Never | 62 | 42 | 43
  Week 80: Wheelchair use: Rarely | 0 | 0 | 0
  Week 80: Wheelchair use: Sometimes | 0 | 0 | 0
  Week 80: Wheelchair use: Often | 0 | 0 | 0
  Week 80: Wheelchair use: Always | 0 | 0 | 0
  Week 80: Device/Utensil to Dress Bathe Eat: number analyzed (Participants) | 62 | 42 | 43
  Week 80: Device/Utensil to Dress Bathe Eat: Never | 62 | 42 | 43
  Week 80: Device/Utensil to Dress Bathe Eat: Rarely | 0 | 0 | 0
  Week 80: Device/Utensil to Dress Bathe Eat: Sometimes | 0 | 0 | 0
  Week 80: Device/Utensil to Dress Bathe Eat: Often | 0 | 0 | 0
  Week 80: Device/Utensil to Dress Bathe Eat: Always | 0 | 0 | 0
  Week 80: Other Aids Or Devices: number analyzed (Participants) | 62 | 42 | 43
  Week 80: Other Aids Or Devices: Never | 62 | 41 | 42
  Week 80: Other Aids Or Devices: Rarely | 0 | 1 | 1
  Week 80: Other Aids Or Devices: Sometimes | 0 | 0 | 0
  Week 80: Other Aids Or Devices: Often | 0 | 0 | 0
  Week 80: Other Aids Or Devices: Always | 0 | 0 | 0

64. Secondary Outcome: Health Care Resource Utilization (HCRU): Number of Participants Who Quit Job Due to Low Back Pain
Description: Low back pain HCRU assessed utilization of healthcare resources during the last 3 months (last 3 months before Baseline [Day 1] visit, weeks 64 and 80 visit, via IRT). Number of participants who answered as "Yes" for quitting job due to low back pain, were evaluated.
Time Frame: Baseline, Weeks 64 and 80
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or placebo matched to tanezumab). Here, 'Number Analyzed' = participants who were evaluable for at specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
Participants
  Baseline | 3 | 2 | 5
  Week 64: number analyzed (Participants) | 91 | 88 | 86
  Week 64 | 1 | 2 | 1
  Week 80: number analyzed (Participants) | 62 | 42 | 43
  Week 80 | 1 | 0 | 0

65. Secondary Outcome: Health Care Resource Utilization (HCRU): Duration Since Quitting Job Due to Low Back Pain
Description: Low back pain HCRU assessed utilization of healthcare resources during the last 3 months (last 3 months before Baseline [Day 1] visit, weeks 64 and 80 visit, via IRT). Domain evaluated was duration (in years) at each specified time point since quitting job due to low back pain.
Time Frame: Baseline, Weeks 64 and 80
Population: ITT population. Not all participants of the ITT population had data collected at each of the time points for this outcome measure. "Overall number of participants analyzed" = participants evaluable for this outcome measure. Additional participants apart from the ones who had responded for quitting job responded to duration since quitting.
Measure: Median (Full Range); unit: years
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 5 | 6 | 6
years
  Baseline: number analyzed (Participants) | 3 | 2 | 5
  Baseline | 1.5 [0.6 to 5.7] | 1.6 [0.3 to 3.0] | 2.5 [0.3 to 10.6]
  Week 64: number analyzed (Participants) | 1 | 4 | 1
  Week 64 | 3.3 [3.3 to 3.3] | 0.7 [0.3 to 1.5] | 0.2 [0.2 to 0.2]
  Week 80: number analyzed (Participants) | 1 | 0 | 0
  Week 80 | 0.1 [0.1 to 0.1] |  |

66. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication Version II (TSQM v II) Scores at Weeks 16 and 56
Description: TSQM v.II: participant rated 11 items questionnaire. Items 1, 2, 7 to 11 were scored as: 1= extremely dissatisfied, 2= very dissatisfied, 3= dissatisfied, 4= somewhat satisfied, 5= satisfied, 6= very satisfied, 7= extremely satisfied. Items 4 to 6 were scored as: 1= extremely dissatisfied, 2= very dissatisfied, 3= somewhat dissatisfied, 4= slightly dissatisfied, 5= not at all dissatisfied. Item 3 was scored as: 0= No, 1= Yes. Four parameters with respect to study medication were evaluated: Effectiveness = ([Item 1+Item 2] - 2 )/12 *100; Side effects = ([Item 4 + Item 5 + Item 6] - 3)/12 *100, if one item is missing then: ([Sum of two completed items]-2]/8 *100; Convenience = ([Item 7 + Item 8 + Item 9] - 3)/18 *100, if one item is missing then: ([Sum of two completed items]-2)/12 *100; Global satisfaction = ([Item 10+Item 11] - 2 ]/12 *100. Each of the 4 parameters had a scale of 0 (no satisfaction) to 100 (best level of satisfaction), higher score = greater satisfaction.
Time Frame: Weeks 16 and 56
Population: ITT population included all randomized participants who received at least one dose of SC study medication (either tanezumab or placebo matched to tanezumab). Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 90 | 88
units on a scale
  Week 16: Effectiveness | 61.41 (21.95) | 61.48 (20.70) | 58.05 (18.97)
  Week 16: Side Effects: number analyzed (Participants) | 6 | 3 | 4
  Week 16: Side Effects | 56.94 (20.01) | 80.56 (19.25) | 68.75 (7.98)
  Week 16: Convenience | 64.79 (17.88) | 66.85 (15.94) | 64.39 (14.31)
  Week 16: Global Satisfaction | 63.41 (20.22) | 62.31 (17.81) | 61.93 (18.17)
  Week 56: Effectiveness: number analyzed (Participants) | 63 | 43 | 43
  Week 56: Effectiveness | 71.30 (20.35) | 71.32 (18.57) | 67.05 (18.63)
  Week 56: Side Effects: number analyzed (Participants) | 0 | 1 | 2
  Week 56: Side Effects |  | 83.33 | 79.17 (5.89)
  Week 56: Convenience: number analyzed (Participants) | 63 | 43 | 43
  Week 56: Convenience | 69.93 (17.78) | 68.86 (16.14) | 68.60 (14.18)
  Week 56: Global Satisfaction: number analyzed (Participants) | 63 | 43 | 43
  Week 56: Global Satisfaction | 72.22 (20.25) | 72.29 (18.61) | 67.44 (15.19)

67. Secondary Outcome: Number of Participants Responding to Patient Reported Treatment Impact Assessment-Modified (mPRTI) at Weeks 16 and 56 for Willingness to Use Study Drug Again
Description: The mPRTI was a self-administered questionnaire containing 4 items to assess participant satisfaction, previous treatment, preference and willingness to continue using the study medication. To assess participants willingness to use study drug again, participants responded using IRT on 5 point Likert scale ranged from 1-5, where, 1= yes, I would definitely want to use the same drug again, 2= I might want to use the same drug again, 3= I am not sure, 4= I might not want to use the same drug again, 5= no, I definitely would not want to use the same drug again. Higher scores indicated lesser willingness to use the study drug.
Time Frame: Weeks 16 and 56
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
Participants
  Week 16: number analyzed (Participants) | 92 | 90 | 88
  Week 16: Yes, definitely want to use the same drug again | 41 | 37 | 40
  Week 16: Might want to use the same drug again | 28 | 27 | 25
  Week 16: I am not sure | 18 | 25 | 21
  Week 16: Might not want to use the same drug again | 3 | 1 | 1
  Week 16: No,definitely wouldn't want to use same drug again | 2 | 0 | 1
  Week 56: number analyzed (Participants) | 63 | 43 | 43
  Week 56: Yes, definitely want to use the same drug again | 34 | 19 | 21
  Week 56: Might want to use the same drug again | 12 | 13 | 15
  Week 56: I am not sure | 16 | 10 | 6
  Week 56: Might not want to use the same drug again | 0 | 1 | 1
  Week 56: No,definitely wouldn't want to use same drug again | 1 | 0 | 0

68. Secondary Outcome: Number of Participants Responding to Patient Reported Treatment Impact Assessment-Modified (mPRTI) at Weeks 16 and 56 for Preference of Study Drug Versus Prior Treatment
Description: The mPRTI was a self-administered questionnaire containing 4 items to assess participant satisfaction, previous treatment, preference and willingness to continue using the study medication. To assess preference to continue using study drug versus previous treatment, participants responded using IRT on 5 point Likert scale from 1-5, where, 1= yes, I definitely prefer drug that I am receiving now, 2= I have a slight preference for drug that I am receiving now, 3= I have no preference either way, 4= I have a slight preference for my previous treatment, 5= No, I definitely prefer my previous treatment. Higher scores indicate lesser preference to use study drug.
Time Frame: Weeks 16 and 56
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
Participants
  Week 16: number analyzed (Participants) | 92 | 90 | 88
  Week 16: Yes, definitely prefer the study drug | 38 | 33 | 31
  Week 16: Slight preference for the study drug | 25 | 26 | 30
  Week 16: No preference either way | 22 | 28 | 23
  Week 16: Slight preference for my previous treatment | 6 | 2 | 3
  Week 16: No, definitely prefer my previous treatment | 1 | 1 | 1
  Week 56: number analyzed (Participants) | 63 | 43 | 43
  Week 56: Yes, definitely prefer the study drug | 33 | 21 | 19
  Week 56: Slight preference for the study drug | 15 | 14 | 16
  Week 56: No preference either way | 13 | 7 | 8
  Week 56: Slight preference for my previous treatment | 0 | 1 | 0
  Week 56: No, definitely prefer my previous treatment | 2 | 0 | 0

69. Primary Outcome: Number of Participants With Abnormal Physical Examination Findings
Description: Physical examination included assessment of general appearance, skin, head, neck, eyes, ears, nose, throat, abdomen, lungs, heart, thyroid, and extremities. Investigator judged abnormality in physical examinations. Only those rows have been reported which had at least 1 participant with abnormality data in any of the reporting arms.
Time Frame: At Screening
Population: Safety analysis population included all participants who were treated with tanezumab or placebo matched to tanezumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
Number analyzed (Participants) | 92 | 93 | 92
Participants
  Skin | 1 | 0 | 3
  Neck | 2 | 1 | 0
  Eyes | 1 | 1 | 1
  Ear | 0 | 1 | 2
  Nose | 0 | 0 | 1
  Extremities | 0 | 1 | 1
  Heart | 2 | 3 | 1

ADVERSE EVENTS:
Time Frame: Baseline up to Week 80
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event.
Arm/Group | Tanezumab 5 mg | Tanezumab 10 mg | Celecoxib
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/93 | 0/92
Serious Adverse Events (participants affected / at risk) | 8/92 | 11/93 | 4/92
Other Adverse Events (participants affected / at risk) | 43/92 | 40/93 | 35/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab 5 mg (N=92) | Tanezumab 10 mg (N=93) | Celecoxib (N=92)
Basedow's disease (Endocrine disorders) | 1 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rapidly progressive osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0
Device dislocation (Product Issues) | 0 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab 5 mg (N=92) | Tanezumab 10 mg (N=93) | Celecoxib (N=92)
Pyrexia (General disorders) | 2 | 2 | 5
Nasopharyngitis (Infections and infestations) | 19 | 19 | 11
Contusion (Injury, poisoning and procedural complications) | 5 | 5 | 3
Fall (Injury, poisoning and procedural complications) | 7 | 6 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 5 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 7 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 2 | 4
Periarthritis (Musculoskeletal and connective tissue disorders) | 6 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 6 | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-07-04): https://cdn.clinicaltrials.gov/large-docs/11/NCT02725411/SAP_000.pdf
  • Study Protocol (2017-09-14): https://cdn.clinicaltrials.gov/large-docs/11/NCT02725411/Prot_001.pdf